### Janssen Research & Development

#### Statistical Analysis Plan

A Randomized, Double-blind, Multicenter, Parallel-Group, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of Aticaprant 10 mg as Adjunctive Therapy in Adult Participants with Major Depressive Disorder (MDD) with Moderate-to-Severe Anhedonia and Inadequate Response to Current Antidepressant Therapy

Protocol 67953964MDD3002; Phase 3

**JNJ-67953964** (aticaprant)

#### **Amendment 3**

Status: Approved

Date: 03 October 2024

Prepared by: Janssen Research & Development, LLC

Document No.: EDMS-RIM-866310; 6.0

Compliance: The study described in this report was performed according to the principles of Good Clinical Practice (GCP).

#### **Confidentiality Statement**

The information provided herein contains Company trade secrets, commercial or financial information that the Company customarily holds close and treats as confidential. The information is being provided under the assurance that the recipient will maintain the confidentiality of the information under applicable statutes, regulations, rules, protective orders or otherwise.

## **TABLE OF CONTENTS**

| TABLE OF C | CONTENTS | 2 |
|---|---|---|
| | VERSION HISTORY | 4 |
| 1. | INTRODUCTION | 7 |
| 1.1. | Objectives and Endpoints | |
| 1.2. | Study Design | |
| 2. | STATISTICAL HYPOTHESES | 13 |
| 3. | SAMPLE SIZE DETERMINATION | |
| 4. | POPULATIONS (ANALYSIS SETS) FOR ANALYSIS | |
| 5. | STATISTICAL ANALYSES | 16 |
| 5.1. | General Considerations | |
| 5.1.1. | Analysis Phases | |
| 5.1.2. | Visit Windows | |
| 5.1.3. | Imputation of Efficacy | |
| 5.1.4. | Country/Territory Pooling Algorithm | |
| 5.2. | Participant Dispositions | |
| 5.3. | Primary Endpoint(s) Analysis | |
| 5.3.1. | Definition | |
| 5.3.2. | Primary Estimand - ROW | |
| 5.3.2.1. | Analysis Methods | |
| 5.3.2.1.1 | Primary Analysis | |
| 5.3.2.1.1. | Sensitivity Analysis | |
| 5.3.2.1.3. | Other Analyses | |
| 5.3.2.1.3.<br>5.4. | | |
| 5.4.<br>5.4.1. | Secondary Endpoint(s) Analysis | |
| 5.4.1.<br>5.4.1.1. | Key Secondary Endpoint | |
| • | Dimensional Anhedonia Rating Scale (DARS) | |
| 5.4.1.1. | Definition | |
| 5.4.1.1.2. | Estimand(s) | |
| 5.4.1.1.3. | Analysis Methods | |
| 5.4.1.1.4. | Other Analyses | |
| 5.4.2. | Other Secondary Endpoint(s) | |
| 5.4.2.1. | Response Based on MADRS Total Score | |
| 5.4.2.1.1. | Definition | |
| 5.4.2.1.2. | Analysis | |
| 5.4.2.2. | Remission Based on MADRS Total Score | |
| 5.4.2.2.1. | Definition | |
| 5.4.2.2.2. | Analysis | |
| 5.4.2.3. | Patient Health Questionnaire - 9 Item (PHQ-9) | |
| 5.4.2.3.1. | Definition | |
| 5.4.2.3.2. | Analysis | |
| 5.4.2.4. | PROMIS Ability to Participate in Social Roles and Activities Short Form 8a (PROMIS Social Roles and Activities Social Roles and Activities Short Form 8a (PROMIS Social Roles and Activities Social Roles and Activities Short Form 8a (PROMIS Social Roles and Activities Social Roles and Activities Social Roles and Activities Short Form 8a (PROMIS Social Roles and Activities Social Roles Activities Social Roles Activities Social Roles Activities Social Roles Activities Social | |
| 54044 | Functioning) | |
| 5.4.2.4.1. | Definition | |
| 5.4.2.4.2. | Analysis | 32 |
| 5.5. | Tertiary/Exploratory Endpoint(s) Analysis | |
| 5.5.1.1. | MADRS-6 | |
| 5.5.1.1.1. | Definition | |
| 5.5.1.1.2. | Analysis | 33 |
| 5.5.1.2. | Snaith-Hamilton Pleasure Scale (SHAPS) | |
| 5.5.1.2.1. | Definition | |
| 5.5.1.2.2. | Analysis | |
| 5.5.1.3. | Clinical Global Impression – Severity (CGI-S) | |
| 5.5.1.3.1. | Definition | |
| 5.5.1.3.2. | Analysis | |
| 5.5.1.4. | Patient Global Impression of Severity (PGI-S) | 34 |

## Statistical Analysis Plan 67953964MDD3002

| 5.5.1.4.2 Analysis .34 5.5.1.5.1 Definition .35 5.5.1.5.1 Definition .35 5.5.1.6.2 Analysis .35 5.5.1.6.1 Definition .35 5.5.1.6.2 Analysis .35 5.5.1.6.1 Definition .36 5.5.1.6.2 Analysis .35 5.5.1.7.1 Quality of Life in Depression Scale (QLDS) .36 5.5.1.7.1 Definition .36 5.5.1.8.1 European Quality of Life (EuroQol) Group, 5 Dimension, 5-Level questionnaire (EQ-5D-5L)36 5.5.1.8.2 Analysis .37 5.5.1.8.3 Safety Analyses .37 5.5.2 Subgroup Analyses .37 5.6.1 Extent of Exposure .38 5.6.1 Extent of Exposure .38 5.6.1 Compliance .38 5.6.2 Adverse Events .38 5.6.3 Actional Safety Assessments .41 5.6.3.1 Clinical Laboratory Tests .41 5.6.3.2 Aiversa and Physical Examination Findings .41 < | 5.5.1.4.1. | Definition | 34 |
|---|---|---|---|
| 5.5.1.5.1 Definition .35 5.5.1.5.2 Analysis .35 5.5.1.6.1 Generalized Anxiety Disorder 7-item Scale (GAD-7) .35 5.5.1.6.2 Analysis .35 5.5.1.7.1 Quality of Life in Depression Scale (QLDS) .36 5.5.1.7.1 Definition .36 5.5.1.8.1 European Quality of Life (EuroQol) Group, 5 Dimension, 5-Level questionnaire (EQ-5D-5L)36 5.5.1.8.1 Definition .36 5.5.1.8.2 Analysis .37 5.5.1.8.1 Definition .38 5.5.1.8.2 Analysis .37 5.6.3 Safety Analyses .37 5.6.3 Safety Analyses .37 5.6.1 Extent of Exposure .38 5.6.2.1 Adverse Events .38 5.6.3.2 Advirage Events .38 5.6.3.3 Additional Safety Assessments .41 5.6.3.4 Other Safety Parameters .41 5.6.3.4 Other Safety Parameters .44 5.6.3.4.2 Other Analyses | 5.5.1.4.2. | Analysis | 34 |
| 5.5.1.6.2 Analysis .35 5.5.1.6. Generalized Anxiety Disorder 7-item Scale (GAD-7) .35 5.5.1.6.1 Definition .35 5.5.1.7. Quality of Life in Depression Scale (QLDS) .36 5.5.1.7.1 Definition .36 5.5.1.8.1 European Quality of Life (EuroQol) Group, 5 Dimension, 5-Level questionnaire (EQ-5D-5L)86 5.5.1.8.2 Luropean Quality of Life (EuroQol) Group, 5 Dimension, 5-Level questionnaire (EQ-5D-5L)86 5.5.1.8.2 Analysis .37 5.5.1.8.2 Subgroup Analyses .37 5.5.1.8.2 Subgroup Analyses .37 5.6.1 Extent of Exposure .38 5.6.1.1 Compliance .38 5.6.2 Adverse Events .38 5.6.3 Additional Safety Assessments .41 5.6.3.1 Clinical Laboratory Tests .41 5.6.3.2 Vital Signs and Physical Examination Findings .41 5.6.3.3 Electrocardiogram .43 5.6.3.4 Columbia Suicide Severity Rating Scale (C-SSRS) .44 5.6.3.4.2 | 5.5.1.5. | Patient Global Impression of Change (PGI-C) | 35 |
| 5.5.1.6.1. Generalized Anxiety Disorder 7-item Scale (GAD-7). .35 5.5.1.6.1. Definition. .35 5.5.1.7. Quality of Life in Depression Scale (QLDS). .36 5.5.1.7.1. Definition. .36 5.5.1.7.2. Analysis. .36 5.5.1.8.1. Definition. .36 5.5.1.8.2. Luopean Quality of Life (EuroQol) Group, 5 Dimension, 5-Level questionnaire (EQ-5D-5L)36 5.5.1.8.2. Analysis. .37 5.5.2. Subgroup Analyses. .37 5.6.2. Analysis. .37 5.6.3. Safety Analyses. .37 5.6.1. Extent of Exposure. .38 5.6.1.1. Compliance. .38 5.6.2. Adverse Events. .38 5.6.3.1. Clinical Laboratory Tests. .41 5.6.3.2. Vital Signs and Physical Examination Findings. .41 5.6.3.4. Other Safety Parameters. .44 5.6.3.4.1. Columbia Suicide Severity Rating Scale (C-SSRS). .44 5.6.3.4.2. Arizona Sexual Experiences Scale ( | 5.5.1.5.1. | Definition | 35 |
| 5.5.1.6.1 Definition .35 5.5.1.6.2 Analysis .35 5.5.1.7.1 Quality of Life in Depression Scale (QLDS) .36 5.5.1.7.2 Analysis .36 5.5.1.8.1 European Quality of Life (EuroQol) Group, 5 Dimension, 5-Level questionnaire (EQ-5D-5L)36 .55.1.8.2 5.5.1.8.2 Analysis .37 5.5.1.8.2 Subgroup Analyses .37 5.6 Safety Analyses .37 5.6.1 Extent of Exposure .38 5.6.1. Extent of Exposure .38 5.6.2 Adverse Events .38 5.6.3. Additional Safety Assessments .41 5.6.3. Additional Safety Assessments .41 5.6.3.1 Clinical Laboratory Tests .41 5.6.3.2 Vital Signs and Physical Examination Findings .41 5.6.3.4. Other Safety Parameters .44 5.6.3.4. Columbia Suicide Severity Rating Scale (C-SSRS) .44 5.6.3.4.1 Columbia Suicide Severity Rating Scale (C-SSRS) .44 5.6.3.4.2 Arizona Sexual Experiences Scale (ASEX) .45 5.6.3. | 5.5.1.5.2. | Analysis | 35 |
| 5.5.1.6.2. Analysis .35 5.5.1.7.1. Definition .36 5.5.1.7.2. Analysis .36 5.5.1.8.1. European Quality of Life (EuroQol) Group, 5 Dimension, 5-Level questionnaire (EQ-5D-5L)36 5.5.1.8.1. Definition .36 5.5.1.8.2. Analysis .37 5.5.2. Subgroup Analyses .37 5.6.1. Extent of Exposure .38 5.6.1. Extent of Exposure .38 5.6.2. Adverse Events .38 5.6.3. Additional Safety Assessments .41 5.6.3.1. Clinical Laboratory Tests .41 5.6.3.2. Vital Signs and Physical Examination Findings .41 5.6.3.3. Clinical Laboratory Tests .41 5.6.3.4. Other Safety Parameters .44 5.6.3.3. Italical Suicide Severity Rating Scale (C-SSRS) .44 5.6.3.4.2. Arizona Sexual Experiences Scale (ASEX) .45 5.6.3.4.2. Physician Withdrawal Checklist 20-item (PWC-20) .46 5.7.1. Pharmacokinetics .46 5.7.2. Biomarkers .46< | 5.5.1.6. | Generalized Anxiety Disorder 7-item Scale (GAD-7) | 35 |
| 5.5.1.7.1 Quality of Life in Depression Scale (QLDS) .36 5.5.1.7.1 Definition .36 5.5.1.8.1 European Quality of Life (EuroQol) Group, 5 Dimension, 5-Level questionnaire (EQ-5D-5L)36 .36 5.5.1.8.1 Definition .36 5.5.1.8.2 Analysis .37 5.5.2 Subgroup Analyses .37 5.6.1 Extent of Exposure .38 5.6.1.1 Compliance .38 5.6.2.1 Adverse Events .38 5.6.3.1 Clinical Laboratory Tests .41 5.6.3.2 Vital Signs and Physical Examination Findings .41 5.6.3.3 Additional Safety Assessments .41 5.6.3.2 Vital Signs and Physical Examination Findings .41 5.6.3.4 Clinical Laboratory Tests .41 5.6.3.4.1 Columbia Suicide Severity Rating Scale (C-SSRS) .44 5.6.3.4.2 Arizona Sexual Experiences Scale (ASEX) .45 5.6.3.4.2.3 Arizona Sexual Experiences Scale (ASEX) .45 5.7.1 Physician Withdrawal Checklist 20-item (PWC-20) <t< td=""><td>5.5.1.6.1.</td><td>Definition</td><td>35</td></t<> | 5.5.1.6.1. | Definition | 35 |
| 5.5.1.7.1 Definition .36 5.5.1.8. European Quality of Life (EuroQoi) Group, 5 Dimension, 5-Level questionnaire (EQ-5D-5L)36 5.5.1.8.1 Definition .36 5.5.1.8.2 Analysis .37 5.5.2 Subgroup Analyses .37 5.6.1 Extent of Exposure .38 5.6.1. Compliance .38 5.6.2. Adverse Events .38 5.6.3. Additional Safety Assessments .41 5.6.3.1 Clinical Laboratory Tests .41 5.6.3.2 Vital Signs and Physical Examination Findings .41 5.6.3.3.2 Vital Signs and Physical Examination Findings .41 5.6.3.4. Other Safety Parameters .44 5.6.3.4.1 Columbia Suicide Severity Rating Scale (C-SSRS) .44 5.6.3.4.2 Arizona Sexual Experiences Scale (ASEX) .45 5.6.3.4.3 Physician Withdrawal Checklist 20-item (PWC-20) .46 5.7.1 Pharmacokinetics .46 5.7.2 Biomarkers .46 5.7.3 Definition of Subgroups .46 6.8 Interim Analyses | 5.5.1.6.2. | Analysis | 35 |
| 5.5.1.7.2 Analysis | 5.5.1.7. | Quality of Life in Depression Scale (QLDS) | 36 |
| 5.5.1.8.1 European Quality of Life (EuroQol) Group, 5 Dimension, 5-Level questionnaire (EQ-5D-5L)36 5.5.1.8.2. Definition 36 5.5.1.8.2. Analysis 37 5.6. Safety Analyses 37 5.6.1. Extent of Exposure 38 5.6.1. Compliance 38 5.6.2. Adverse Events 38 5.6.3. Additional Safety Assessments 41 5.6.3.1. Clinical Laboratory Tests 41 5.6.3.2. Vital Signs and Physical Examination Findings 41 5.6.3.3. Electrocardiogram 43 5.6.3.4. Other Safety Parameters 44 5.6.3.4. Other Safety Parameters 44 5.6.3.4.2. Arizona Sexual Experiences Scale (ASEX) 45 5.6.3.4.2. Arizona Withdrawal Checklist 20-item (PWC-20) 46 5.7.1. Pharmacokinetics 46 5.7.2. Biomarkers 46 5.7.3. Definition of Subgroups 46 5.8. Interim Analyses 48 5.8. | 5.5.1.7.1. | Definition | 36 |
| 5.5.1.8.1 Definition .36 5.5.1.8.2 Analysis .37 5.5.2 Subgroup Analyses .37 5.6.1 Extent of Exposure .38 5.6.1. Extent of Exposure .38 5.6.1. Compliance .38 5.6.2 Adverse Events .38 5.6.3. Additional Safety Assessments .41 5.6.3.1 Clinical Laboratory Tests .41 5.6.3.2 Vital Signs and Physical Examination Findings .41 5.6.3.3. Electrocardiogram .43 5.6.3.4 Other Safety Parameters .44 5.6.3.4.1 Columbia Suicide Severity Rating Scale (C-SSRS) .44 5.6.3.4.2 Arizona Sexual Experiences Scale (ASEX) .45 5.6.3.4.3 Physician Withdrawal Checklist 20-item (PWC-20) .46 5.7 Other Analyses .46 5.7.1 Pharmacokinetics .46 5.7.2 Biomarkers .46 5.7.3 Definition of Subgroups .46 5.8.1 Interim Analyses .48 5.8.1 Independent Data M | 5.5.1.7.2. | | |
| 5.5.1. Analysis .37 5.5.2. Subgroup Analyses .37 5.6. Safety Analyses .37 5.6.1. Extent of Exposure .38 5.6.1. Compliance .38 5.6.2. Adverse Events .38 5.6.3. Additional Safety Assessments .41 5.6.3.1. Clinical Laboratory Tests .41 5.6.3.2. Vital Signs and Physical Examination Findings .41 5.6.3.3. Electrocardiogram .43 5.6.3.4. Other Safety Parameters .44 5.6.3.4.1. Columbia Suicide Severity Rating Scale (C-SSRS) .44 5.6.3.4.2. Arizona Sexual Experiences Scale (ASEX) .45 5.6.3.4.3. Physician Withdrawal Checklist 20-item (PWC-20) .46 5.7. Other Analyses .46 5.7.1. Pharmacokinetics .46 5.7.2. Biomarkers .46 5.7.3. Definition of Subgroups .46 5.8. Interim Analyses .48 5.8.1. Independent Data Monitoring Committee (IDMC) .48 5.8. | 5.5.1.8. | European Quality of Life (EuroQoI) Group, 5 Dimension, 5-Level questionnaire (EQ-5D-5 | 5L)36 |
| 5.5.2. Subgroup Analyses .37 5.6. Safety Analyses .37 5.6.1. Extent of Exposure .38 5.6.2. Adverse Events .38 5.6.3. Additional Safety Assessments .41 5.6.3.1. Clinical Laboratory Tests .41 5.6.3.2. Vital Signs and Physical Examination Findings .41 5.6.3.3. Electrocardiogram .43 5.6.3.4. Other Safety Parameters .44 5.6.3.4.1. Columbia Suicide Severity Rating Scale (C-SSRS) .44 5.6.3.4.2. Arizona Sexual Experiences Scale (ASEX) .45 5.6.3.4.3. Physician Withdrawal Checklist 20-item (PWC-20) .46 5.7. Other Analyses .46 5.7.1. Pharmacokinetics .46 5.7.2. Biomarkers .46 5.7.3. Definition of Subgroups .46 5.8. Interim Analyses .48 5.8. Interim Analyses .48 6.1. Appendix 1 List of Abbreviations .48 6.2. Appendix 2 Changes to Protocol-Planned Analyses .51 </td <td>5.5.1.8.1.</td> <td>Definition</td> <td>36</td> | 5.5.1.8.1. | Definition | 36 |
| 56. Safety Analyses .37 5.6.1. Extent of Exposure .38 5.6.1. Compliance .38 5.6.2. Adverse Events .38 5.6.3. Additional Safety Assessments .41 5.6.3.1. Clinical Laboratory Tests .41 5.6.3.2. Vital Signs and Physical Examination Findings .41 5.6.3.3. Electrocardiogram .43 5.6.3.4. Other Safety Parameters .44 5.6.3.4. Columbia Suicide Severity Rating Scale (C-SSRS) .44 5.6.3.4.2. Arizona Sexual Experiences Scale (ASEX) .45 5.7. Other Analyses .46 5.7.1. Pharmacokinetics .46 5.7.2. Biomarkers .46 5.7.3. Definition of Subgroups .46 5.8.1. Independent Data Monitoring Committee (IDMC) .48 6. SUPPORTING DOCUMENTATION .48 6.1. Appendix 1 List of Abbreviations .48 6.2. Appendix 2 Changes to Protocol-Planned Analyses .51 | 5.5.1.8.2. | Analysis | 37 |
| 5.6.1. Extent of Exposure .38 5.6.1. Compliance .38 5.6.2. Adverse Events .38 5.6.3. Additional Safety Assessments .41 5.6.3.1. Clinical Laboratory Tests .41 5.6.3.2. Vital Signs and Physical Examination Findings .41 5.6.3.3. Electrocardiogram .43 5.6.3.4. Other Safety Parameters .44 5.6.3.4.1. Columbia Suicide Severity Rating Scale (C-SSRS) .44 5.6.3.4.2. Arizona Sexual Experiences Scale (ASEX) .45 5.6.3.4.3. Physician Withdrawal Checklist 20-item (PWC-20) .46 5.7.1. Pharmacokinetics .46 5.7.2. Biomarkers .46 5.7.3. Definition of Subgroups .46 5.8. Interim Analyses .48 5.8.1. Independent Data Monitoring Committee (IDMC) .48 6. SUPPORTING DOCUMENTATION .48 6.1. Appendix 1 List of Abbreviations .48 6.2. Appendix 2 Changes to Protocol-Planned Analyses .51 6.3. Appendix 3 Demo | 5.5.2. | Subgroup Analyses | 37 |
| 5.6.1.1 Compliance .38 5.6.2. Adverse Events .38 5.6.3. Additional Safety Assessments .41 5.6.3.1. Clinical Laboratory Tests .41 5.6.3.2. Vital Signs and Physical Examination Findings .41 5.6.3.4. Other Safety Parameters .43 5.6.3.4.1. Columbia Suicide Severity Rating Scale (C-SSRS) .44 5.6.3.4.2. Arizona Sexual Experiences Scale (ASEX) .45 5.6.3.4.3. Physician Withdrawal Checklist 20-item (PWC-20) .46 5.7. Other Analyses .46 5.7.1. Pharmacokinetics .46 5.7.2. Biomarkers .46 5.7.3. Definition of Subgroups .46 5.8. Interim Analyses .48 5.8.1. Independent Data Monitoring Committee (IDMC) .48 6. SUPPORTING DOCUMENTATION .48 6.1. Appendix 1 List of Abbreviations .48 6.2. Appendix 2 Changes to Protocol-Planned Analyses .51 6.3. Appendix 3 Demographics and Baseline Characteristics .52 6.4. | 5.6. | Safety Analyses | 37 |
| 5.6.1.1 Compliance .38 5.6.2. Adverse Events .38 5.6.3. Additional Safety Assessments .41 5.6.3.1. Clinical Laboratory Tests .41 5.6.3.2. Vital Signs and Physical Examination Findings .41 5.6.3.4. Other Safety Parameters .43 5.6.3.4.1. Columbia Suicide Severity Rating Scale (C-SSRS) .44 5.6.3.4.2. Arizona Sexual Experiences Scale (ASEX) .45 5.6.3.4.3. Physician Withdrawal Checklist 20-item (PWC-20) .46 5.7. Other Analyses .46 5.7.1. Pharmacokinetics .46 5.7.2. Biomarkers .46 5.7.3. Definition of Subgroups .46 5.8. Interim Analyses .48 5.8.1. Independent Data Monitoring Committee (IDMC) .48 6. SUPPORTING DOCUMENTATION .48 6.1. Appendix 1 List of Abbreviations .48 6.2. Appendix 2 Changes to Protocol-Planned Analyses .51 6.3. Appendix 3 Demographics and Baseline Characteristics .52 6.4. | 5.6.1. | Extent of Exposure | 38 |
| 5.6.3. Additional Safety Assessments .41 5.6.3.1. Clinical Laboratory Tests .41 5.6.3.2. Vital Signs and Physical Examination Findings .41 5.6.3.3. Electrocardiogram .43 5.6.3.4. Other Safety Parameters .44 5.6.3.4.1. Columbia Suicide Severity Rating Scale (C-SSRS) .44 5.6.3.4.2. Arizona Sexual Experiences Scale (ASEX) .45 5.6.3.4.3. Physician Withdrawal Checklist 20-item (PWC-20) .46 5.7. Other Analyses .46 5.7.1. Pharmacokinetics .46 5.7.2. Biomarkers .46 5.7.3. Definition of Subgroups .46 5.8. Interim Analyses .48 5.8.1. Independent Data Monitoring Committee (IDMC) .48 6.8.1. Appendix 1 List of Abbreviations .48 6.1. Appendix 2 Changes to Protocol-Planned Analyses .51 6.3. Appendix 3 Demographics and Baseline Characteristics .52 6.4. Appendix 5 Prior and Concomitant Medications .54 6.5. Appendix 6 Medications of Special Interest | 5.6.1.1. | | |
| 5.6.3.1. Clinical Laboratory Tests. .41 5.6.3.2. Vital Signs and Physical Examination Findings .41 5.6.3.3. Electrocardiogram .43 5.6.3.4. Other Safety Parameters .44 5.6.3.4.1. Columbia Suicide Severity Rating Scale (C-SSRS). .44 5.6.3.4.2. Arizona Sexual Experiences Scale (ASEX). .45 5.6.3.4.3. Physician Withdrawal Checklist 20-item (PWC-20). .46 5.7. Other Analyses. .46 5.7.1. Pharmacokinetics. .46 5.7.2. Biomarkers. .46 5.7.3. Definition of Subgroups. .46 5.8.1. Independent Data Monitoring Committee (IDMC). .48 5.8.1. Independent Data Monitoring Committee (IDMC). .48 6.1. Appendix 1 List of Abbreviations. .48 6.2. Appendix 2 Changes to Protocol-Planned Analyses. .51 6.3. Appendix 3 Demographics and Baseline Characteristics. .52 6.4. Appendix 4 Protocol Deviations. .54 6.5. Appendix 5 Prior and Concomittant Medications. .56 6.6. Appe | 5.6.2. | Adverse Events | 38 |
| 5.6.3.2. Vital Signs and Physical Examination Findings | 5.6.3. | Additional Safety Assessments | 41 |
| 5.6.3.3. Electrocardiogram .43 5.6.3.4. Other Safety Parameters. .44 5.6.3.4.1. Columbia Suicide Severity Rating Scale (C-SSRS). .44 5.6.3.4.2. Arizona Sexual Experiences Scale (ASEX). .45 5.6.3.4.3. Physician Withdrawal Checklist 20-item (PWC-20). .46 5.7. Other Analyses. .46 5.7.1. Pharmacokinetics. .46 5.7.2. Biomarkers. .46 5.7.3. Definition of Subgroups. .46 5.8. Interim Analyses. .48 5.8.1. Independent Data Monitoring Committee (IDMC). .48 6.1. Appendix 1 List of Abbreviations .48 6.1. Appendix 1 List of Abbreviations .48 6.2. Appendix 2 Changes to Protocol-Planned Analyses. .51 6.3. Appendix 3 Demographics and Baseline Characteristics .52 6.4. Appendix 4 Protocol Deviations .54 6.5. Appendix 5 Prior and Concomitant Medications .55 6.6. Appendix 6 Medications of Special Interest .56 6.7. Appendix 7 Conversion of Raw Score to T-Sco | 5.6.3.1. | Clinical Laboratory Tests | 41 |
| 5.6.3.4. Other Safety Parameters. .44 5.6.3.4.1. Columbia Suicide Severity Rating Scale (C-SSRS) .44 5.6.3.4.2. Arizona Sexual Experiences Scale (ASEX) .45 5.6.3.4.3. Physician Withdrawal Checklist 20-item (PWC-20) .46 5.7. Other Analyses .46 5.7.1. Pharmacokinetics .46 5.7.2. Biomarkers .46 5.8. Interim Analyses .46 5.8.1. Independent Data Monitoring Committee (IDMC) .48 6. SUPPORTING DOCUMENTATION .48 6.1. Appendix 1 List of Abbreviations .48 6.2. Appendix 2 Changes to Protocol-Planned Analyses .51 6.3. Appendix 2 Changes to Protocol-Planned Analyses .51 6.4. Appendix 3 Demographics and Baseline Characteristics .52 6.4. Appendix 5 Prior and Concomitant Medications .52 6.5. Appendix 5 Prior and Concomitant Medications .55 6.6. Appendix 6 Medications of Special Interest .56 6.7. Appendix 8 Criteria for Treatment-emergent Markedly Abnormal Laboratory Values .58 | 5.6.3.2. | Vital Signs and Physical Examination Findings | 41 |
| 5.6.3.4.1. Columbia Suicide Severity Rating Scale (C-SSRS) | 5.6.3.3. | Electrocardiogram | 43 |
| 5.6.3.4.2. Arizona Sexual Experiences Scale (ASEX) 45 5.6.3.4.3. Physician Withdrawal Checklist 20-item (PWC-20) 46 5.7. Other Analyses 46 5.7.1. Pharmacokinetics 46 5.7.2. Biomarkers 46 5.7.3. Definition of Subgroups 46 5.8. Interim Analyses 48 5.8.1. Independent Data Monitoring Committee (IDMC) 48 6. SUPPORTING DOCUMENTATION 48 6.1. Appendix 1 List of Abbreviations 48 6.2. Appendix 2 Changes to Protocol-Planned Analyses 51 6.3. Appendix 3 Demographics and Baseline Characteristics 52 6.4. Appendix 4 Protocol Deviations 54 6.5. Appendix 5 Prior and Concomitant Medications 55 6.6. Appendix 6 Medications of Special Interest 56 6.7. Appendix 6 Medications of Special Interest 56 6.8. Appendix 7 Conversion of Raw Score to T-Score for PROMIS 57 6.8. Appendix 8 Criteria for Treatment-emergent Markedly Abnormal Laboratory Values 58 6.9. Appendi | 5.6.3.4. | Other Safety Parameters | 44 |
| 5.6.3.4.3. Physician Withdrawal Checklist 20-İtem (PWC-20) 46 5.7. Other Analyses 46 5.7.1. Pharmacokinetics 46 5.7.2. Biomarkers 46 5.7.3. Definition of Subgroups 46 5.8. Interim Analyses 48 5.8.1. Independent Data Monitoring Committee (IDMC) 48 6. SUPPORTING DOCUMENTATION 48 6.1. Appendix 1 List of Abbreviations 48 6.2. Appendix 2 Changes to Protocol-Planned Analyses 51 6.3. Appendix 3 Demographics and Baseline Characteristics 52 6.4. Appendix 4 Protocol Deviations 54 6.5. Appendix 5 Prior and Concomitant Medications 55 6.6. Appendix 6 Medications of Special Interest 56 6.7. Appendix 7 Conversion of Raw Score to T-Score for PROMIS 57 6.8. Appendix 8 Criteria for Treatment-emergent Markedly Abnormal Laboratory Values 58 6.9. Appendix 9 Analyses for Assessing and Mitigating the Impact of COVID- 19 on Study 60 6.10. Appendix 10 Delta Adjustment Multiple Imputation 61 | 5.6.3.4.1. | Columbia Suicide Severity Rating Scale (C-SSRS) | 44 |
| 5.7. Other Analyses 46 5.7.1. Pharmacokinetics 46 5.7.2. Biomarkers 46 5.7.3. Definition of Subgroups 48 5.8. Interim Analyses 48 5.8.1. Independent Data Monitoring Committee (IDMC) 48 6. SUPPORTING DOCUMENTATION 48 6.1. Appendix 1 List of Abbreviations 48 6.2. Appendix 2 Changes to Protocol-Planned Analyses 51 6.3. Appendix 3 Demographics and Baseline Characteristics 52 6.4. Appendix 4 Protocol Deviations 54 6.5. Appendix 4 Protocol Deviations 54 6.5. Appendix 5 Prior and Concomitant Medications 55 6.6. Appendix 6 Medications of Special Interest 56 6.7. Appendix 7 Conversion of Raw Score to T-Score for PROMIS 57 6.8. Appendix 8 Criteria for Treatment-emergent Markedly Abnormal Laboratory Values 58 6.9. Appendix 9 Analyses for Assessing and Mitigating the Impact of COVID- 19 on Study 60 6.10. Appendix 10 Delta Adjustment Multiple Imputation 61 6.11. </td <td>5.6.3.4.2.</td> <td>Arizona Sexual Experiences Scale (ASEX)</td> <td>45</td> | 5.6.3.4.2. | Arizona Sexual Experiences Scale (ASEX) | 45 |
| 5.7.1. Pharmacokinetics 46 5.7.2. Biomarkers 46 5.7.3. Definition of Subgroups 46 5.8. Interim Analyses 48 5.8.1. Independent Data Monitoring Committee (IDMC) 48 6. SUPPORTING DOCUMENTATION 48 6.1. Appendix 1 List of Abbreviations 48 6.2. Appendix 2 Changes to Protocol-Planned Analyses 51 6.3. Appendix 2 Demographics and Baseline Characteristics 52 6.4. Appendix 3 Demographics and Baseline Characteristics 52 6.4. Appendix 4 Protocol Deviations 54 6.5. Appendix 5 Prior and Concomitant Medications 55 6.6. Appendix 6 Medications of Special Interest 56 6.7. Appendix 7 Conversion of Raw Score to T-Score for PROMIS 57 6.8. Appendix 8 Criteria for Treatment-emergent Markedly Abnormal Laboratory Values 58 6.9. Appendix 9 Analyses for Assessing and Mitigating the Impact of COVID- 19 on Study 0utcome 60 6.10. Appendix 10 Delta Adjustment Multiple Imputation 61 6.12. Appendix | 5.6.3.4.3. | Physician Withdrawal Checklist 20-item (PWC-20) | 46 |
| 5.7.2. Biomarkers | 5.7. | Other Analyses | 46 |
| 5.7.3. Definition of Subgroups | 5.7.1. | Pharmacokinetics | 46 |
| 5.8. Interim Analyses | 5.7.2. | Biomarkers | 46 |
| 5.8.1.Independent Data Monitoring Committee (IDMC)486.SUPPORTING DOCUMENTATION486.1.Appendix 1 List of Abbreviations486.2.Appendix 2 Changes to Protocol-Planned Analyses516.3.Appendix 3 Demographics and Baseline Characteristics526.4.Appendix 4 Protocol Deviations546.5.Appendix 5 Prior and Concomitant Medications556.6.Appendix 6 Medications of Special Interest566.7.Appendix 7 Conversion of Raw Score to T-Score for PROMIS576.8.Appendix 8 Criteria for Treatment-emergent Markedly Abnormal Laboratory Values586.9.Appendix 9 Analyses for Assessing and Mitigating the Impact of COVID- 19 on Study<br>Outcome606.10.Appendix 10 Delta Adjustment Multiple Imputation616.11.Appendix 11 AE Suggested to Abuse Potential (PTs)636.12.Appendix 12 Spaghetti Plot of MADRS Change Over Time (Study 67953964MDD2001)646.13.Appendix 13 Quality Tolerance Limits (QTLs)656.14.Appendix 14 Scoring of QLDS items66 | 5.7.3. | Definition of Subgroups | 46 |
| 5.8.1.Independent Data Monitoring Committee (IDMC)486.SUPPORTING DOCUMENTATION486.1.Appendix 1 List of Abbreviations486.2.Appendix 2 Changes to Protocol-Planned Analyses516.3.Appendix 3 Demographics and Baseline Characteristics526.4.Appendix 4 Protocol Deviations546.5.Appendix 5 Prior and Concomitant Medications556.6.Appendix 6 Medications of Special Interest566.7.Appendix 7 Conversion of Raw Score to T-Score for PROMIS576.8.Appendix 8 Criteria for Treatment-emergent Markedly Abnormal Laboratory Values586.9.Appendix 9 Analyses for Assessing and Mitigating the Impact of COVID- 19 on Study<br>Outcome606.10.Appendix 10 Delta Adjustment Multiple Imputation616.11.Appendix 11 AE Suggested to Abuse Potential (PTs)636.12.Appendix 12 Spaghetti Plot of MADRS Change Over Time (Study 67953964MDD2001)646.13.Appendix 13 Quality Tolerance Limits (QTLs)656.14.Appendix 14 Scoring of QLDS items66 | 5.8. | Interim Analyses | 48 |
| 6.1.Appendix 1 List of Abbreviations486.2.Appendix 2 Changes to Protocol-Planned Analyses516.3.Appendix 3 Demographics and Baseline Characteristics526.4.Appendix 4 Protocol Deviations546.5.Appendix 5 Prior and Concomitant Medications556.6.Appendix 6 Medications of Special Interest566.7.Appendix 7 Conversion of Raw Score to T-Score for PROMIS576.8.Appendix 8 Criteria for Treatment-emergent Markedly Abnormal Laboratory Values586.9.Appendix 9 Analyses for Assessing and Mitigating the Impact of COVID- 19 on Study Outcome606.10.Appendix 10 Delta Adjustment Multiple Imputation616.11.Appendix 11 AE Suggested to Abuse Potential (PTs)636.12.Appendix 12 Spaghetti Plot of MADRS Change Over Time (Study 67953964MDD2001)646.13.Appendix 13 Quality Tolerance Limits (QTLs)656.14.Appendix 14 Scoring of QLDS items66 | 5.8.1. | Independent Data Monitoring Committee (IDMC) | 48 |
| 6.2.Appendix 2 Changes to Protocol-Planned Analyses516.3.Appendix 3 Demographics and Baseline Characteristics526.4.Appendix 4 Protocol Deviations546.5.Appendix 5 Prior and Concomitant Medications556.6.Appendix 6 Medications of Special Interest566.7.Appendix 7 Conversion of Raw Score to T-Score for PROMIS576.8.Appendix 8 Criteria for Treatment-emergent Markedly Abnormal Laboratory Values586.9.Appendix 9 Analyses for Assessing and Mitigating the Impact of COVID- 19 on Study<br>Outcome606.10.Appendix 10 Delta Adjustment Multiple Imputation616.11.Appendix 11 AE Suggested to Abuse Potential (PTs)636.12.Appendix 12 Spaghetti Plot of MADRS Change Over Time (Study 67953964MDD2001)646.13.Appendix 13 Quality Tolerance Limits (QTLs)656.14.Appendix 14 Scoring of QLDS items66 | 6. | SUPPORTING DOCUMENTATION | 48 |
| 6.2.Appendix 2 Changes to Protocol-Planned Analyses516.3.Appendix 3 Demographics and Baseline Characteristics526.4.Appendix 4 Protocol Deviations546.5.Appendix 5 Prior and Concomitant Medications556.6.Appendix 6 Medications of Special Interest566.7.Appendix 7 Conversion of Raw Score to T-Score for PROMIS576.8.Appendix 8 Criteria for Treatment-emergent Markedly Abnormal Laboratory Values586.9.Appendix 9 Analyses for Assessing and Mitigating the Impact of COVID- 19 on Study<br>Outcome606.10.Appendix 10 Delta Adjustment Multiple Imputation616.11.Appendix 11 AE Suggested to Abuse Potential (PTs)636.12.Appendix 12 Spaghetti Plot of MADRS Change Over Time (Study 67953964MDD2001)646.13.Appendix 13 Quality Tolerance Limits (QTLs)656.14.Appendix 14 Scoring of QLDS items66 | 6.1. | Appendix 1 List of Abbreviations | 48 |
| 6.4. Appendix 4 Protocol Deviations | 6.2. | Appendix 2 Changes to Protocol-Planned Analyses | 51 |
| 6.5. Appendix 5 Prior and Concomitant Medications | 6.3. | Appendix 3 Demographics and Baseline Characteristics | 52 |
| 6.6. Appendix 6 Medications of Special Interest | 6.4. | Appendix 4 Protocol Deviations | 54 |
| 6.7. Appendix 7 Conversion of Raw Score to T-Score for PROMIS | 6.5. | | |
| 6.8. Appendix 8 Criteria for Treatment-emergent Markedly Abnormal Laboratory Values | 6.6. | Appendix 6 Medications of Special Interest | 56 |
| 6.9. Appendix 9 Analyses for Assessing and Mitigating the Impact of COVID- 19 on Study Outcome 60 6.10. Appendix 10 Delta Adjustment Multiple Imputation 61 6.11. Appendix 11 AE Suggested to Abuse Potential (PTs) 63 6.12. Appendix 12 Spaghetti Plot of MADRS Change Over Time (Study 67953964MDD2001) 64 6.13. Appendix 13 Quality Tolerance Limits (QTLs) 65 6.14. Appendix 14 Scoring of QLDS items 66 | 6.7. | | |
| Outcome | 6.8. | Appendix 8 Criteria for Treatment-emergent Markedly Abnormal Laboratory Values | 58 |
| 6.10. Appendix 10 Delta Adjustment Multiple Imputation | 6.9. | Appendix 9 Analyses for Assessing and Mitigating the Impact of COVID- 19 on Study | |
| 6.11. Appendix 11 AE Suggested to Abuse Potential (PTs) | | Outcome | 60 |
| 6.12. Appendix 12 Spaghetti Plot of MADRS Change Over Time (Study 67953964MDD2001)64 6.13. Appendix 13 Quality Tolerance Limits (QTLs) | 6.10. | | |
| 6.12. Appendix 12 Spaghetti Plot of MADRS Change Over Time (Study 67953964MDD2001)64 6.13. Appendix 13 Quality Tolerance Limits (QTLs) | 6.11. | Appendix 11 AE Suggested to Abuse Potential (PTs) | 63 |
| 6.13. Appendix 13 Quality Tolerance Limits (QTLs) | | Appendix 12 Spaghetti Plot of MADRS Change Over Time (Study 67953964MDD2001). | 64 |
| | | Appendix 13 Quality Tolerance Limits (QTLs) | 65 |
| | | Appendix 14 Scoring of QLDS items | |

## **VERSION HISTORY**

Table - SAP Version History Summary

| SAP<br>Version | Approval<br>Date | Change | Rationale |
|---|---|---|---|
| 6.0 | 04Oct<br>2024 | Removed Appendix 14 and Appendix 15<br>Statistical Analysis Plan for Japan/China-<br>specific protocol | Details about the analysis sets and statistical analyses for these countries/territories will be described in separate analysis plans specific to Japan (if needed) and China. |
| 5.0 | 09Aug<br>2024 | Minor typo fix | |
| 4.0 | 08Aug<br>2024 | Section 5.4.1.1.4 Mediation analysis: updated the direction of the arrow in the mediation analysis figure | To clarify |
| | | Section 6.1 Appendix 1 List of Abbreviations: updated the contents for MDD_WOANH_MS and MDD_WOANH_MS | To be consistent with analysis set definition |
| | | Section 6.3: removed "MDD Anhedonia status" from the psychiatric history table Section 6.14, 6.15: Replaced FAS_ANH-with newly defined non-enriched populations | The information will be presented in the table of summary of analysis sets Replaced the FAS_ANH- analysis set with the newly defined non-enriched populations for the statistical analysis plan for the Japan and China |
| | | Section 7: deleted citations that are not referenced in the main body of the document | For consistency |
| 3.0 | 31Jul<br>2024 | Sections 1, 1.1, 1.2, 3, 5.1.4: replaced MDD ANH- with Non-PAP | Non-PAP more accurately reflects the population, i.e., subjects who are not in the primary analysis set. |
| | | Section 4, 5.1, 5.6.1, 5.6.1.1, 6.3: Replaced FAS_ANH- with newly defined non-enriched populations | The FAS_ANH- population will not be analyzed as a separate group as a portion of this population includes participants with prominent anhedonia Hence, replaced the analysis set with the newly defined non-enriched populations. |
| | | Sections 5.1.4, 5.4.2.3.2: Removed MDD ANH- | Same as above |
| | | Section 5.1.4 Pooling Algorithm: Further details added for clarity | To clarify |
| | | Section 5.3.2.1.1 Primary Analysis: Algorithms for MMRM with unstructured and structured covariance implemented based on the FDA's instruction. | Based on FDA comments |
| | | Sections 5.3.2.1.3, 5.4.1.1.4: Added additional analyses for the newly defined non-enriched populations. | The All MDD group contains non_PAP, the group of participants that does not reflect the non-enriched population of interest. |
| | | Removed interaction test for the All MDD group. Deleted analysis of additional subpopulations | Formal statistical analyses will not be performed due to insufficient sample size in non-enriched subgroups. |

Statistical Analysis Plan 67953964MDD3002

| SAP<br>Version | Approval | Change | Dationals |
|---|---|---|---|
| version | Date | Change Section 5.4.1.1.4 baseline MADRS added | Rationale To help address the potential mediator- |
| | | in ANCOVA mediation analysis for the | outcome confounding. |
| | | change in DARS total score. | cuttome comountaing. |
| | | Section 5.6.2: Added additional AE | To better characterize the safety profile of |
| | | summaries | aticaprant |
| | | Section 5.6.3.1 Laboratory Tests: further | To clarify. |
| | | detail added for hepatic abnormality. | |
| | | | Shift table is not needed for interpretation |
| | | Deleted shift table. | of safety profile as aticaprant use is not associated with metabolic effects and there |
| | | | are no metabolic related endpoints. |
| | | Section 5.6.3.4.2 ASEX: Subgroup of | It is more appropriate to explore the |
| | | responder status by MADRS at Day 43 | subgroups at baseline. |
| | | removed | sucgroups at ouseffice. |
| | | Section 5.7.3: New subgroups added | To better characterize the treatment effect |
| | | - | in various sub-groups |
| | | Section 6.3, Table 7 demographic variables | To better characterize the study population |
| | | and Table 8 psychiatric history: | |
| | | demographic and baseline variables added | T. 1 'C |
| | | Throughout the document: Added additional information for clarity | To clarify |
| 2.0 | 26 Feb | Updated "Subjects" to "participants" | To be consistent with the template |
| 2.0 | 2024 | throughout the document | To be consistent with the template |
| | | Replaced "actual value" with "observed | To use a more accurate term |
| | | value" throughout the document | |
| | | Section 1.1 Objectives and Endpoints: | Updated to align with protocol amendment |
| | | minor updates to descriptions for endpoints | 1. |
| | | Section 3 Updated the sample size | To be consistent with the modification to |
| | | determination section | the criteria that define MDD ANH+. |
| | | Section 5 General Considerations: Updated the stratification criteria based on MDD | To clarify the new stratification criteria for MDD AHN status |
| | | ANH status in the interactive web response | IVIDD ATIN Status |
| | | system (IWRS). | |
| | | Section 5.1.1 Added "Start and end dates | To clarify |
| | | for the follow-up phase are only defined for | |
| | | participants who continue into the follow- | |
| | | up phase." | |
| | | Table 1 Merged scales with the same | To simplify the table |
| | | assessment schedules together | T. 1 'C14' 1' 4 4 |
| | | Section 5.3.2 Updates made to primary estimand -ROW | To clarify population and intercurrent events |
| | | Section 5.3.2.1 Updated delta adjustment | To clarify delta adjustment and provide |
| | | analysis and added an additional sensitivity | further sensitivity analysis |
| | | analysis for MMRM with an additional | |
| | | fixed effect factor of MDD ANH status | |
| | | (MDDANH1, MDDANH2). | |
| | | Section 5.3.2.1.3 Other analysis: removed | To simplify analyses planed. |
| | | forest plot for LS mean change of MARDS | To Update SHAPS cut off and address |
| | | for FAS_ANH+, FAS_ANH- and | FDA request |
| | | FAS_All. Updated the sub-population planed for | |
| | | FAS All, CCI and | |
| | | added sub-population based on MADRS | |
| | | item 8 | |

#### Statistical Analysis Plan 67953964MDD3002

| SAP | Approval | | atistical Analysis Plan 67953964MDD3002 |
|---|---|---|---|
| Version | Date | Change | Rationale |
| | | Section 5.3.2.1.3 Removed mediation | To clarify the interest of the mediation |
| | | analysis of change of MADRS mediated by | analysis is the evaluation of the effect of |
| | | change of DARS | aticaprant on anhedonia that is independent |
| | | | from the effect on depression. |
| | | Section 5.5.1.2, 5.5.1.5 and 5.5.1.6 Updated | To clarify |
| | | descriptions of SHAPS, PGI-C, and GAD-7 | |
| | | Section 5.5.1.8 Updated analysis part of | To clarify |
| | | EQ-5-D | |
| | | Section 5.6.1 Extent of Exposure Updated | To clarify |
| | | the definition of total number of dosing | |
| | | days | |
| | | Section 5.6.1.1 Updated the calculation of | |
| | | compliance for current AD | |
| | | Added "DB phase" for safety analysis in | To clarify the analysis will only be |
| | | Section 5.6.2 and 5.6.3 | performed in DB phase |
| | | Section 5.6.2 Added additional analyses for | To clarify the details of analyses for AESI |
| | | AESI | |
| | | Added "RR interval" to Table 6 | To clarify the additional parameter included |
| | | Section 5.6.3.4.1 Added a listing for C- | To clarify additional analysis |
| | | SSRS | m '1 11'0' 1 1 ' |
| | | Section 5.6.4.3.2 Added subgroup analyses for ASEX | To provide additional analysis |
| | | Removed Analysis for "menstrual Cycle | Excluded analysis with limited value in a |
| | | Tracking" | short term study |
| | | Section 5.7.3 Updated the definition of | To clarify the subgroups that will be |
| | | subgroup "Race", merged categories with | explored |
| | | few subjects | |
| | | Updated Appendix 9 | To clarify when COVID-19 related analysis |
| | | | will be performed |
| | | Appendix 14 and 15 Updates made to the | To clarify and be consistent with primary |
| | | population of primary estimand -Japan and | estimand - ROW |
| | | China | |
| | | Other minor changes in | To clarify |
| | | wording/terminology made throughout the | |
| | | document. | |
| 1 | 20 Mar | Not Applicable | Initial release |
| | 2023 | | |

#### 1. INTRODUCTION

This statistical analysis plan (SAP) contains definitions of analysis sets, derived variables, and statistical methods for all planned analyses for study 67953964MDD3002.

The 'MDD ANH-' population that is referenced in the protocol has been renamed in the SAP as non-primary analysis population or 'non-PAP' to more accurately reflect the population, as some subjects in this population had prominent anhedonia

## 1.1. Objectives and Endpoints

This is a randomized, double-blind, multicenter, parallel-group, placebo-controlled study to evaluate the efficacy, safety, and tolerability of aticaprant 10 mg as adjunctive therapy in adult participants with major depressive disorder (MDD) with moderate-to-severe anhedonia and inadequate response to current antidepressant therapy.

#### **OBJECTIVES AND ENDPOINTS**

| Objectives | Endpoints |
|---|---|
| Primary | • |
| • To evaluate the efficacy of aticaprant 10 m compared with placebo as adjunctive therapy to a antidepressant in improving depressive symptom in adult participants with MDD with moderate-to severe anhedonia (ANH+) who have had a inadequate response to current antidepressar therapy with an SSRI or SNRI. | pre-randomization, and hereafter referred to as 'baseline') to Day 43 in the Montgomery-Åsberg Depression Rating Scale (MADRS) total score |
| Key Secondary | |
| To evaluate the efficacy of adjunctive aticaprar 10 mg compared with placebo in improvin anhedonia in adult participants with MDD ANH who have had an inadequate response to currer antidepressant therapy with an SSRI or SNRI | Dimensional Anhedonia Rating Scale (DARS) total score |
| Other Secondary | |
| To evaluate the efficacy of aticaprant 10 mg compared antidepressant in adult participants with MDD ANH+ antidepressant therapy (SSRI or SNRI) on the following Depressive symptoms (clinician-reported) | who have had an inadequate response to the current |
| | MADRS total score. |
| Response of depressive symptoms (clinician-<br>reported) | • Proportion of responders on depressive symptoms scale, defined as a ≥50% improvement in MADRS total score from baseline to Day 43. |
| • Remission of depressive symptoms (clinician-reported) | • Proportion of participants with remission of depressive symptoms, defined as a MADRS total score ≤10 at Day 43. |

| Objectives | Endpoints |
|---|---|
| Symptoms of depression (patient-reported) | Change from baseline to Day 43 in Patient |
| Symptoms of depression (patient-reported) | Health Questionnaire, 9-Item (PHQ-9) total score. |
| Anhedonia symptoms (patient-reported) | Change from baseline over time in DARS total score. |
| | • Change from baseline over time in the PHQ-9 anhedonia-specific item (PHQ-9, item 1). |
| | • Proportion of participants with a score less than 2 in the PHQ-9 anhedonia-specific item (PHQ-9, item 1) at Day 43. |
| Social functioning (patient-reported) | Change from baseline over time in the<br>Patient-Reported Outcomes Measurement<br>Information System (PROMIS) Short Form<br>v2.0 – Ability to Participate in Social Roles<br>and Activities - 8a (PROMIS-APS 8a) |
| Safety | |
| All participants - Safety will be assessed for all MDD p | articipants (adult and elderly). |
| • To assess the safety and tolerability of aticaprant 10 mg as adjunctive therapy to an antidepressant | AEs, including AEs of special interest (AESI) |
| (SSRI or SNRI) in all MDD participants (adult and elderly) in short-term treatment compared | Vital signs |
| with placebo. | • 12-lead ECG |
| | Laboratory parameters |
| | Weight/Body Mass Index (BMI) |
| | Suicidality assessment using the C-SSRS |
| | • Withdrawal symptoms assessment using the physician Withdrawal Checklist 20-items (PWC 20). |
| | Proportion of participants with clinically relevant sexual dysfunction over time in the Arizona Sexual Experiences Scale (ASEX) score. |
| Exploratory | 1 |
| To assess the efficacy of aticaprant 10 mg compared wit (SSRI or SNRI) in adult participants with MDD ANH+ (adult and elderly participants with MDD ANH+ and n their current antidepressant therapy on the following: | (PAP), adult non-PAP, and all MDD participants |
| Depressive symptoms (clinician and patient-reported). | Change from baseline over time in the MADRS total score (applicable to adult non-PAP and All MDD). |
| | • Change from baseline over time in the MADRS-6 score. |

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

Statistical Analysis Plan 67953964MDD3002

| Objectives | Endpoints |
|---|---|
| | Change from baseline over time in PHQ-9 total score. |
| Anhedonia symptoms (patient-reported) | Change from baseline over time in DARS total score (applicable to adult non-PAP and All MDD). |
| | Change from baseline over time in the subscales of the DARS (hobbies/pastimes, food/drink, social activities, and sensory experiences). |
| | Change from baseline in the Snaith-<br>Hamilton Pleasure Scale (SHAPS) over<br>time. |
| | • DARS improvement response at Day 43 (increase in DARS total score ≥ meaningful change threshold [or range of thresholds] determined by anchor-based analyses of blinded interim data, as indicated in Section 5.8) |
| Severity of depressive symptoms (clinician- and patient- reported) | Change from baseline over time in the<br>Clinical Global Impression-Severity (CGI-S) score |
| | <ul> <li>Change from baseline over time in the<br/>symptoms of depression as assessed using<br/>the Patient Global Impression of Severity<br/>(PGI-S) for depression.</li> </ul> |
| Severity of anhedonia symptoms (patient-reported) | Change from baseline over time in anhedonia symptoms using the PGI-S for anhedonia. |
| | • Score at Day 43 in anhedonia symptoms using the PGI-C for anhedonia. |
| Health-related quality of life (patient-reported) | Change from baseline over time in health-<br>related quality of life EQ visual analogue<br>scale (EQ-VAS) and health status, as<br>assessed by the European Quality of Life, 5<br>Dimension, 5Level (EQ-5D-5L)<br>questionnaire. |
| | Change from baseline over time in health-<br>related quality of life as assessed by the<br>Quality of Life in Depression Scale<br>(QLDS). |
| Anxiety symptoms (patient-reported) | Change from baseline to Day 43 in symptoms of anxiety using the Generalized Anxiety Disorder 7-item Scale (GAD-7). |

| | Statistical Alialysis Flail 0/955904NIDD5002 |
|---|---|
| Objectives | Endpoints |
| Clinical Pharmacology Assessments | |

#### Clinical Pharmacology Assessments

- To assess the pharmacokinetics of aticaprant (10 mg) in participants with MDD when used as adjunctive treatment.
- To assess the exposure-response relationship of aticaprant and MADRS in participants with MDD.
- To assess the exposure-response relationship of aticaprant and selected adverse events.

#### **Biomarker Signatures**

- To confirm the diagnostic biomarker signature identified in Study 67953964MDD3001 which might be predictive of clinical improvement on depression symptoms and anhedonia upon treatment with aticaprant.
- To explore genetic and other factors that may influence the efficacy, pharmacokinetics, safety, or tolerability of aticaprant.
- To confirm the diagnostic value of biosignature identified in Study 67953964MDD3001 to predict treatment response.
- Change from baseline to Day 43 in MADRS total score in defined biosignature positive participants and respective biosignature negative participants.

#### Digital Biomarkers

- To evaluate the association between digital biomarkers at baseline (derived from speech, video, and Reward Learning Task [RLT]) and treatment response.
- To evaluate the correlation of digital biomarkers with measures of anhedonia and other depression characteristics, and Biomarker Signature defined subgroup.
- To evaluate the change of exploratory digital endpoint (for example, RLT from block 1 to block 2 or from block 1 to block 3, learning rate, and reward sensitivity [ie, baseline to Day 43]).

## 1.2. Study Design

This is a multicenter, randomized, double-blind, parallel-group, placebo-controlled study to assess the efficacy, safety and tolerability of adjunctive aticaprant 10 mg in adult participants (18 to 64 years of age, inclusive) who have major depressive disorder (MDD) with moderate-to-severe anhedonia (MDD ANH+, also referred to as the Primary Analysis Population [PAP]), adult participants who do not qualify for MDD ANH+ (non-PAP), and elderly participants (65 to 74 years of age, inclusive) with MDD (ANH+ and non-PAP). All participants must have had an inadequate response to a selective serotonin reuptake inhibitor (SSRI) or serotonin-norepinephrine reuptake inhibitor (SNRI) in the current depressive episode.

In addition, PK, pharmacogenomics, and biomarkers will also be evaluated.

This study will consist of the following phases:

- Screening Phase (evaluate eligibility): up to 30 days prior to first dose administration.
- Double-blind (DB) Treatment Phase: 43 days.
- Follow-up Phase: up to 14 days.

Figure 1: Schematic Overview of the Study



Approximately 538 participants (430 adult and 108 elderly) will be randomized. The adult MDD ANH+ population randomized to aticaprant 10 mg or placebo will be included in the primary and key secondary analysis.

Additionally, approximately 118 participants from China and/or 54 participants from Japan (if participating) will be enrolled in the study.

All participants will continue to take their current SSRI or SNRI antidepressant therapy (at the same dose and at approximately the same time of the day) throughout the study.

Abbreviations: SSRI = selective serotonin reuptake inhibitor; SNRI = serotonin norepinephrine reuptake inhibitor.

Participants will be randomized in a 1:1 ratio to receive aticaprant at 10 mg or placebo for 42 days. The study intervention will be administered orally as 2 film-coated tablets to be taken together, once daily, around the same time and preferably in the morning.

The study population will include participants who meet Diagnostic and Statistical Manual of Mental Disorders-5th Edition (DSM-5) diagnostic criteria for recurrent or single episode MDD, without psychotic features, based upon clinical assessment and confirmed by the Structured Clinical Interview for DSM-5 Axis I Disorders - Clinical Trials Version (SCID-CT). Participants 65 years of age or older must have had the first onset of depression prior to 55 years of age. Eligible participants must have a 17-item Hamilton Depression Rating Scale (HDRS-17) total score ≥20 at the first and second screening interviews with no greater than 20% improvement from the first to the second independent HDRS-17 assessments at screening. Moreover, all participants must have had an inadequate response to at least 1 oral antidepressant treatment (SSRI or SNRI), administered at an adequate dose (therapeutic dose per MGH ATRQ) and duration (at least 6 weeks) in the current depressive episode. An inadequate response is defined as <50% reduction in depressive symptom severity but with some improvement (>0%; i.e., there may be minimal to moderate symptomatic improvement since the initiation of treatment, but some of the initial symptoms are still present, troubling to the participant and affecting behavior and function) as assessed by the MGH-ATRQ. The inadequate response must include the participant's current SSRI/SNRI treatment.

All participants will continue their current SSRI/SNRI antidepressant at the same dose without change and taken approximately around the same time of the day as prior to entering the Screening and DB Treatment Phase.

Participants are considered to have completed the DB Treatment Phase of the study if they have completed the Day 43 visit of the DB Treatment Phase, including the MADRS assessment at the end of the 6-week DB Treatment Phase (i.e., Day 43 MADRS), and have not discontinued study intervention early during the DB Treatment Phase.

Participants who have completed the DB Treatment Phase (Day 43) and were compliant to the study intervention may be eligible to participate in a separate 52-week open-label long-term safety study 67953964MDD3003. The investigator and the participant will determine, based on efficacy and tolerability of the DB treatment, whether it is in the best interest of the participant to continue treatment in the open-label long-term safety study. The decision to enroll in the 67953964MDD3003 study or enter the Follow-up Phase will be documented in the electronic case report form (eCRF). Participants who complete the DB Treatment Phase, are eligible and decide to roll-over to the open-label long-term safety study are not expected to complete the Follow-up Phase.

Participants who complete the DB Treatment Phase will be considered to have completed the study if they roll over to Study 67953964MDD3003 or complete the Follow-up Visit, including the MADRS, DARS, and PWC-20 assessments at this visit. If a participant enters the open-label safety study, the Follow-up Visit will not be conducted.

Participants who discontinue study intervention in the DB Treatment Phase will be considered to have completed the study if they completed the Follow-up Phase, including the MADRS, DARS, and PWC-20 assessments at this visit.

Participants who discontinue study intervention early (i.e., prior to completion of Day 43 visit) or who are non-compliant to the study intervention (i.e., have missed either 4 or more consecutive doses of study intervention or a total of 8 or more doses during the DB Treatment Phase) will not be eligible to participate in the open-label safety study.

Participants who discontinue study intervention during the DB Treatment Phase and participants who completed of the DB Treatment Phase who are not rolling-over to the open-label long-term safety study (67953964MDD3003) will complete the End-of-Treatment (EOT)/Early Withdrawal (EW) visit and will then enter the Follow-up Phase of the study.

No study intervention will be administered during the Follow up Phase; further clinical/standard of care for the treatment of depression will be arranged by the study investigator and/or participant's treating physician, and changes to current antidepressant treatment are permitted in this study phase.

The worldwide COVID-19 pandemic may impact the conduct of clinical studies due to the challenges from quarantines, site closures, travel limitations, and other considerations if site personnel or study participants become potentially exposed to or infected with COVID-19. To assure the safety of study participants, maintain compliance with Good Clinical Practice (GCP), and minimize risks to study integrity, if necessary, in consultation with the sponsor, the method of assessments may be changed (e.g., paper assessments replaced by electronic assessments and vice versa). In addition, site visits may be replaced with telephone, internet-based video-conferencing applications, or home visits by qualified healthcare professionals (HCP). Rating scales/safety assessments can continue to be administered via video teleconferencing (MADRS) or phone (other assessments). Every effort should be made to complete the MADRS assessment via video teleconferencing and within the scheduled timeframe; if this cannot occur, the sponsor medical monitor or delegate should be contacted for direction. Normal procedures, as detailed in this protocol, will be resumed as soon as possible thereafter. For participants who receive an approved or authorized vaccine, it is recommended that this occurs at least 5 days prior to the start of dosing, or once randomized at least 5 days prior to the next scheduled visit.

An Independent Data Monitoring Committee (IDMC) will be commissioned to periodically review safety data for this study.

#### 2. STATISTICAL HYPOTHESES

This study is designed to show that the treatment effect in improving depressive symptoms (as measured by change from baseline on Day 43 in MADRS total score) of aticaprant 10 mg as an adjunctive MDD treatment is superior to placebo in adult participants with MDD ANH+.

If  $\mu_T$  is the mean change in MADRS total score for the aticaprant 10 mg group and  $\mu_P$  is the mean change in MADRS total score for the placebo group, then the hypothesis can be written as follows:

$$H_0: \mu_T - \mu_P \ge 0 \text{ vs}$$
  
 $H_1: \mu_T - \mu_P < 0$ 

Superiority can be concluded if the two-sided p-value for the testing of the hypothesis above is less than 0.05 (2-sided) and the direction is consistent with the alternative hypothesis.

#### 3. SAMPLE SIZE DETERMINATION

Approximately 538 participants, including adult (18 to 64 years of age, inclusive) and elderly (65 to 74 years of age, inclusive) will be randomized in this study.

Participants entering the DB Treatment phase will be randomized in a 1:1 ratio to adjunctive placebo, and adjunctive aticaprant 10 mg. A minimum of 324 adult participants with MDD ANH+ and approximately 106 adult non-PAP will be randomized.

Assuming an effect size of 0.38 for the change in MADRS total score, and a 1-sided significance level of 0.025 (equivalently, 2-sided 0.05), this sample size of 324 adult participants with MDD ANH+ will provide approximately 88% power for the comparison between adjunctive aticaprant 10 mg and adjunctive placebo for the primary efficacy endpoint (in adult participants with MDD ANH+), accounting for a dropout rate of approximately 15%.

The effect size used in the sample size calculation was based on the results of Study 67953964MDD2001 where the effect size was 0.39 (mean difference between treatment groups of -3.4 and a pooled standard deviation of 8.72) for the change from baseline to Day 43 in MADRS total score for the relevant study population, and clinical judgment.

It is expected that approximately 108 elderly participants (65 to 74 years of age, inclusive) will be randomized in the study. This subset of participants will be analyzed as an exploratory evaluation and will not be included in the primary analysis set.

Additionally, approximately 118 participants from China will participate in the study. In the event Japan participates in the study, approximately 54 participants will be enrolled in this country/territory. The details are described in the respective country/territory-specific amendments to the protocol.

**Note**: The sample size assumptions are based on the criteria that define MDD ANH+. These criteria have been modified from the protocol, which are documented in the protocol addendum. Based on the results from the Phase 2 study using the new criteria, the study is powered for the original planned number of 324 participants with MDD ANH+. The table below provides the differences between the protocol and the SAP.

| | Phase 3 study | y | Results from Study 67953964MDD2001 | | |
|---|---|---|---|---|---|
| Document | Assumed Effect<br>Size | Power | Effect size | Mean treatment<br>difference | Pooled standard deviation |
| Protocol | 0.4 | 90% | 0.45 | -4.1 | 8.98 |
| SAP | 0.38 | 88% | 0.39 | -3.4 | 8.72 |

## 4. POPULATIONS (ANALYSIS SETS) FOR ANALYSIS

The following analysis sets are defined for the participants enrolled in rest of world (ROW i.e., countries/territories other than China and Japan).

| Population | Description |
|---|---|
| All Participants | All participants in ROW who sign the informed consent form (ICF) |
| Randomized | All participants in ROW who were randomized in the study |
| Full Analysis Set | All adult randomized participants in ROW with MDD ANH+ who take at least 1 |
| (ANH+) (FAS_ANH+) | dose of study intervention. This is the primary analysis population for the |
| | primary and key secondary efficacy endpoints. |
| MDD_WOANH_S | Adult randomized participants in ROW with CCI |
| Analysis Set who take at least 1 dose of study intervention. | |
| MDD_WOANH_MS | WOANH_MS Adult randomized participants in ROW with CCI |
| Analysis Set | who take at least 1 dose of study |
| | intervention. |
| Full Analysis Set (All) All randomized participants (adult and elderly) in ROW with MDD ANH+ of | |
| (FAS All) | non-PAP who take at least 1 dose of study intervention |
| Safety Analysis Set | All randomized participants (adults and elderly) in ROW who take at least 1 |
| | dose of study intervention. |
| Follow-up Analysis Set | All randomized participants in ROW who entered the follow-up phase after the |
| | double-blind treatment phase |
| | he treatment effect in participants without anhedonia, analyses will be conducted |
| for the MDD WOANH | S and MDD WOANH MS analysis sets as noted in the relevant sections below. |

Due to Good Clinical Practice (GCP) issues, participants enrolled in the Scarpino site will be included in the randomized analysis set, but not in the efficacy and safety analysis sets. Patient profiles will be provided for these participants.

#### 5. STATISTICAL ANALYSES

#### 5.1. General Considerations

As indicated in Section 3 the criteria defining MDD ANH+ were modified while the study was ongoing. Hence the stratification criteria based on MDD ANH status was also modified in the interactive web response system (IWRS). While the original stratification consisted of two strata – MDD ANH+ and MDD ANH-, the modified stratification scheme consists of three strata – MDDANH1

Details about the modification to the criteria are presented in the addendum to the protocol which is blinded to the study sites. The mapping of the different strata from the 2 schemes is presented in Figure 2.

Figure 2: MDD ANH Stratification in IWRS – Mapping of MDD ANH Strata between Original and Modified



For participants who were randomized under the original scheme, participants from the MDD ANH+ stratum will be classified under MDDANH1, and those from the stratum called MDD ANH- stratum will be classified into MDDANH2 and MDDANH3. For all the analyses described in this document the primary population of interest, i.e., adult participants with MDD with moderate-to-severe anhedonia (referred to as 'MDD ANH+' in the protocol), will include adult participants belonging to MDDANH1 and MDDANH2. Participants in the MDDANH3 stratum will be termed as the non-PAP group.

It is possible that the enrollment in Japan (if participating) and/or China may take significantly longer than the ROW. Therefore, so as not to delay ROW submissions, data from Japan and China will only be combined with the global data for local registration in the respective countries/territories. Analyses of efficacy data from the ROW will be used for submissions outside of Japan and China. Details about the analysis sets and statistical analyses for these countries/territories will be described in a separate document specific to Japan (if needed) and China.

The assessment of the primary and secondary (key and other) endpoints will be conducted on the FAS\_ANH+, which includes adult (not elderly) participants with MDD ANH+ who were randomized to aticaprant 10 mg or placebo and took at least 1 dose of study intervention. The exploratory endpoints will be analyzed in adult participants with MDD ANH+ (FAS\_ANH+), and all MDD participants (FAS\_All: adult and elderly participants with MDD ANH+ and non-PAP). As the non-PAP group also consists of participants with moderate-to-severe anhedonia exploratory endpoints described in the protocol will not be analyzed for this population. Similar classification will be applied to elderly participants who are included in FAS\_All.

The primary efficacy endpoint is the change in MADRS total score from baseline to Day 43 in adult participants with MDD ANH+. The key secondary endpoint is the change in DARS total score from baseline to Day 43 in this group of study participants.

## 5.1.1. Analysis Phases

#### **Double-Blind Treatment Phase**

The analysis reference start date of the double-blind treatment phase (DB phase start date) is the date of the first dose of double-blind study intervention. The analysis reference end date of the double-blind treatment phase (DB phase end date) is the maximum of the date of the last visit in the double-blind treatment phase and date of completion or early withdrawal from the double-blind treatment phase.

For randomized participants who did not receive any study intervention in the double-blind treatment phase, both analysis reference start and end dates are missing for the double-blind treatment phase.

#### Follow-up Phase

Start and end dates for the follow-up phase are only defined for participants who continue into the follow-up phase. The analysis reference start date of the follow-up phase (follow-up phase start date) is the day after the reference end date for the double-blind treatment phase. The analysis reference end date of the follow-up phase (follow-up phase end date) is the maximum of the date of the last visit in the follow-up phase and trial disposition.

#### 5.1.2. Visit Windows

As participants do not always adhere to the protocol visit schedule, the following rules are applied to assign actual visits to analysis visits. Listed below are the visit windows and the target days for each visit. The reference day is Study Day 1. If a participant has 2 or more actual visits in a visit window, the visit closest to the target day will be used as the protocol visit for that visit window. The other additional visit(s) will not be used in the summaries or analyses, but they can be used for determination of clinically important endpoints. If 2 actual visits are equidistant from the target day within a visit window, the later visit is used.

All assignments will be made in chronological order. Once a visit date is assigned to a visit window, it will no longer be used for a later time point except for the endpoint. Listed below (Table 1) are the analysis visit windows and the target days for each visit defined in the protocol.

#### Table 1- Visit Windows

| Parameter | Analysis<br>Phase | Scheduled<br>Visit Number | Time<br>Interval | Time Interval<br>(Day)* | Target<br>Time<br>Point |
|---|---|---|---|---|---|
| MADRS, | DB | 2.1 | Baseline (DB) | ( <b>Day</b> ) | 1 |
| DARS, | - | 2.3 | Day 15 | 2 to 22 | 15 |
| CGI-S, | - | 2.5 | Day 13 Day 29 | 23 to 36 | 29 |
| PGI-S anhedonia, | - | 2.7 | Day 43 | 37 to End of DB | 43 |
| PHQ-9, | - | DB final visit | Endpoint (DB) | 2 to End of DB | 43 |
| PGI-S depression, | | | | 2 to End of DB | |
| PROMIS SF 8a,<br>EQ-5D-5L | FU | 3.1 | Follow-up | End of DB + 1 to<br>End of FU | 7-14 |
| QLDS, | DB | 2.1 | Baseline (DB) | <=1 | 1 |
| ASEX | | 2.5 | Day 29 | 2 to 36 | 29 |
| | | 2.7 | Day 43 | 37 to End of DB | 43 |
| | | DB final visit | Endpoint (DB) | 2 to End of DB | |
| SHAPS | SCR | 1.1 | Screening | <1 | |
| | DB | 2.1 | Baseline (DB) | <=1 | 1 |
| | | 2.3 | Day 15 | 2 to 22 | 15 |
| | | 2.5 | Day 29 | 23 to 36 | 29 |
| | | 2.7 | Day 43 | 37 to End of DB | 43 |
| | | DB final visit | Endpoint (DB) | 2 to End of DB | |
| GAD-7 | DB | 2.1 | Baseline (DB) | <=1 | 1 |
| | | 2.7 | Day 43 | 2 to End of DB | 43 |
| | | DB final visit | Endpoint (DB) | 2 to End of DB | |
| PGI-C anhedonia | DB | 2.7 | Day 43 | 1 to End of DB | 43 |
| | | DB final visit | Endpoint (DB) | 1 to End of DB | |
| PWC-20 | DB | 2.7 | Day 43 | 1 to End of DB | 43 |
| | | DB final visit | Endpoint (DB) | 1 to End of DB | |
| | FU | 3.1 | Follow-up | End of DB + 1 to | 7-14 |
| Vital Signs | SCR | 1.1 | Screening | <1 | |
| | DB | 2.1 | Baseline (DB) | <=1 | 1 |
| | | 2.3 | Day 15 | 2 to 22 | 15 |
| | | 2.5 | Day 29 | 23 to 36 | 29 |
| | | 2.7 | Day 43 | 37 to End of DB | 43 |
| | | DB final visit | Endpoint (DB) | 2 to End of DB | |
| | FU | 3.1 | Follow-up | End of DB + 1 to<br>End of FU | 7-14 |
| ECG | SCR | 1.1 | Screening | <1 | |
| | DB | 2.1 | Baseline (DB) Day 1: Postdose | <=1/ predose | 1 |
| | | 2.5 | Day 29: Predose<br>Day 29: Postdose | 2 to 36 | 29 |
| | | 2.7 | Day 43 | 37 to End of DB | 43 |
| | | DB final visit | Endpoint (DB) | 2 to End of DB | |
| Hematology, | SCR | 1.1 | Screening | <1 | |
| Chemistry | DB | 2.1 | Baseline (DB) | <=1 | 1 |
| Urinalysis | F | 2.7 | Day 43 | 2 to End of DB | 43 |
| | Ī | DB final visit | Endpoint (DB) | 2 to End of DB | |
| C-SSRS | SCR | 1.1 | Screening | <1 | |
| ļ | DB | 2.1 | Baseline (DB) | <=1 | 1 |
| | F | 2.2 | Day 8 | 2 to 11 | 8 |
| | F | 2.3 | Day 15 | 12 to 18 | 15 |
| | ļ | 2.4 | Day 22 | 19 to 25 | 22 |
| | ļ | 2.5 | Day 29 | 26 to 32 | 29 |
| | - | 2.6 | Day 36 | 33 to 39 | 36 |

| | | 2.7 | Day 43 | 40 to End of DB | 43 |
|------------|-----|----------------|---------------|------------------|------|
| | | DB final visit | Endpoint (DB) | 2 to End of DB | |
| | FU | 3.1 | Follow-up | End of DB + 1 to | 7-14 |
| Weight/BMI | SCR | 1.1 | Screening | <1 | |
| | DB | 2.1 | Baseline (DB) | <=1 | 1 |
| | | 2.7 | Day 43 | 2 to End of DB | 43 |
| | | DB final visit | Endpoint (DB) | 2 to End of DB | |
| | FU | 3.1 | Follow-up | End of DB + 1 to | 7-14 |
| | | | | End of FU | |

<sup>\*</sup>Relative to the first day of the DB phase. For the follow-up phase, time interval is relative to the first day of the follow-up phase, and Day 11 in this phase will be considered as target day if there are multiple assessments.

Relative day: (event date – analysis phase start date + 1) for an event occurring on or after the analysis phase start date; (event date – analysis phase start date) for an event prior to the analysis phase start date.

Baseline (DB) is the last observation prior to or on the start date of DB phase. Endpoint (DB) is the last observation in the DB phase.

#### 5.1.3. Imputation of Efficacy

Imputation for missing data in the primary and key secondary endpoint (MADRS and DARS) will include the following methods (Table 2).

**Table 2: Imputation of Missing Efficacy Data** 

| Imputation | Method/Rule |
|---|---|
| Multiple Imputation (MI) method | Delta Adjustment |
| Non-Responder | Participants with missing values will be imputed as non-responders for analyses that use imputed data. |
| Non-Remitter | Participants with missing values will be imputed as non-remitters for analyses that use imputed data. |

Imputation of total scores will be performed for the efficacy scales as shown in Table 3 below. If the number of items with missing scores is greater than the maximum number of items that can be missing (as presented in the table), the total score will be missing.

For the remaining efficacy assessments which require adding multiple item scores, the total score will be missing if any item score is missing.

**Table 3: Imputation of Total Score for Efficacy Scales** 

| Efficacy Scale | Total<br>Number of<br>Items | Maximum Number<br>of Items That Can<br>Be Missing | Formula for Total Score |
|---|---|---|---|
| MADRS | 10 | 1 | Sum of non-missing item scores * (10 |
| | | | / number of non-missing items) |
| QLDS | 34 | 6 | Sum of non-missing item scores * (34 |
| | | | / number of non-missing items) |

# 5.1.4. Country/Territory Pooling Algorithm

Pooling will be conducted if a sufficient number of participants are not randomized to a country/territory. If necessary, the countries/territories with fewer than 4 randomized participants will be combined for the purpose of analysis within each region (North America, Europe, South America, Asia, and Other). These countries/territories will be ordered according to the total number of participants. The pooling will be carried out sequentially beginning with the smallest countries/territories until the number of participants in the pooled analysis countries/territories is 4 or more. The size of any pooled analysis countries/territories should be as large as possible and not be larger than the size of the largest country/territory in the region. If the number of small countries/territories is large, and one pooled analysis country/territory cannot include all small countries/territories, then the second (or more) pooled analysis country/territory will be formed after the first one is filled with as many small countries/territories as possible. Pooled countries/territories as described are called analysis countries/territories and will be used in the analyses as country/territory effect.

Pooling will be conducted in adult participants with MDD ANH+. The same procedure will be applied for all MDD participants (adult and elderly participants with MDD ANH+ and non-PAP).

## 5.2. Participant Dispositions

The number of screened participants and reason for screen failures will be summarized overall.

The number of participants in the following disposition categories will be summarized throughout the study by intervention group and overall for the all randomized, FAS All and FAS ANH+:

- Participants randomized
- Participants who received study intervention
- Participants who completed, discontinued and reasons for discontinuation of study intervention during double-blind phase
- Participants who completed, terminated and reasons for discontinuation of study
- Intercurrent events in the double-blind phase

The number of participants in each analysis set will be provided.

Listings of participants will be provided for the following categories:

- Participants who discontinued double-blind study intervention
- Participants who were unblinded during the study period
- Participants who were randomized yet did not receive study intervention.

If deemed necessary, additional analyses of disposition data for assessing and mitigating the impact of COVID-19 on study outcome will be conducted as presented in Appendix 9.

## 5.3. Primary Endpoint(s) Analysis

#### 5.3.1. Definition

The primary efficacy endpoint is the change from baseline in MADRS total score at Day 43 in FAS ANH+.

The MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant intervention. The scale consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms). Higher scores represent a more severe condition. The MADRS evaluates reported sadness, apparent sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. The test exhibits high inter-rater reliability. The typical recall period for the MADRS is 7 days.

The MADRS total score is the sum of scores from individual question items at a given time point, and ranges from 0 to 60. Higher scores represent a more severe condition. Imputation of total score is presented in Section 5.1.3.

Negative changes in MADRS total score indicate improvement.

The sections below describe the primary and sensitivity analyses performed for each primary and supplementary estimand.

## 5.3.2. Primary Estimand - ROW

This estimand is defined to address the primary objective when the study intervention is taken as directed.

**Primary Trial Objective**: To evaluate the efficacy of aticaprant 10 mg compared with placebo as adjunctive therapy to an antidepressant in improving depressive symptoms in adult participants with MDD ANH+ who have had an inadequate response to current antidepressant therapy with an SSRI or SNRI.

**Estimand Scientific Question of Interest**: What is the antidepressant benefit from aticaprant 10 mg versus placebo as adjunctive treatment to a SSRI or SNRI in adult participants with MDD ANH+, who have had an inadequate response to current antidepressant therapy with an SSRI or SNRI based on the change from baseline in MADRS total score if the participants take study intervention as directed?

This estimand is defined by the following 5 components:

#### **Study Intervention:**

- Experimental: Aticaprant 10 mg as an adjunctive treatment to SSRI or SNRI
- Control: Placebo as an adjunctive treatment to SSRI or SNRI

**Population**: Adult patients (18 to 64 years of age, inclusive) in ROW with a diagnosis of MDD ANH+ who have had an inadequate response to current antidepressant therapy with an SSRI/SNRI.

Variable: Change in MADRS total score from baseline to Day 43

Summary Measure: Difference in intervention means

Intercurrent events and their corresponding strategies:

| | Intercurrent Events | Name of Strategy for Addressing<br>Intercurrent Events and Its Description |
|---|---|---|
| 1. | Discontinuation of study intervention only | Hypothetical strategy: as if the intercurrent event had not occurred |
| 2. | Discontinuation of both study intervention and current antidepressant | Hypothetical strategy: see above |
| 3. | Switch of study intervention only (ie, initiation of another antidepressant after discontinuation of study intervention) | Hypothetical strategy: see above |
| 4. | Switch of current antidepressant therapy only | Hypothetical strategy: see above |
| 5. | Switch of study intervention and current antidepressant therapy | Hypothetical strategy: see above |

For participants experiencing multiple intercurrent events at the same time or switching study intervention and/or current antidepressant therapy after discontinuation of study intervention and/or current antidepressant therapy before/on the end of DB phase, intercurrent events in categories 3-5 will override the rest. For example, if a patient starts a new antidepressant medication the day after taking the last dose of their study intervention/current antidepressant therapy, this intercurrent event will be considered a switch of study intervention/current antidepressant therapy, and not a discontinuation. However, if more than one day passes between the last dose of their study intervention/current antidepressant therapy and the first dose of the new antidepressant medication, this situation will be considered a discontinuation of study intervention/current antidepressant therapy intercurrent event followed by a switch of antidepressant medication intercurrent event.

For all intercurrent events, data collected beyond 1 week from the occurrence of the event (or the first event in participants with multiple ICEs) including the data from the EOT/EW visit will be excluded from the analysis. No additional intercurrent events will be assigned beyond 1 week from the occurrence of the first intercurrent event.

Rationale for including data collected within 1 week from the occurrence of the intercurrent event: Given the weekly schedule of data collection (either via a telephone contact, or at a site visit) the expectation is that it could take up to a week for the participants to schedule the EOT/EW visit. This window of data collection post-ICE aligns with aticaprant's mean half-life (t½) of 21.3 to 38.5 hours (IB Aticaprant 2022). Additionally, for the ICEs of switch to a new antidepressant treatment the time to an onset of initial effect for the most commonly prescribed antidepressants is typically at least 2 to 4 weeks (Khin, 2013; Yang, 2013).

## 5.3.2.1. Analysis Methods

#### 5.3.2.1.1. Primary Analysis

The change from baseline in MADRS total score will be analyzed by a Mixed-Effect Model for Repeated Measures (MMRM) based on observed data. The fixed terms included in the model will be intervention group (aticaprant 10 mg and placebo), country/territory, time, and time-by intervention interaction, and the baseline score as a covariate. The within-subject covariance between visits will be estimated via an unstructured variance-covariance matrix. The Kenward-Roger method will be used for approximating the denominator degrees of freedom. In case of convergence problems, with the default Newton Raphson algorithm, alternative approaches will be tried in the following order before using a structured variance-covariance matrix: Fisher scoring algorithm, and factor analysis structure. If the convergence issues persist with the unstructured variance-covariance matrix, alternative variance-covariance structures will be tried in the following order, with the first structure that converges being used in the analysis: heterogeneous Toeplitz, standard Toeplitz, and AR(1) with separate subject random effect. A robust sandwich variance estimator will be used if a structured covariance matrix is implemented. Comparison between aticaprant 10 mg and placebo at Day 43 will be performed using the appropriate contrast. The least square (LS) mean (+/-SE) change from baseline and the difference of LS means (95% CI) will be presented over time.

Descriptive statistics of the observed values and the change from baseline to each time point in the double-blind and follow-up phases will be presented for MADRS total score by intervention group.

Justification of MMRM using MAR assumption: The discontinuation rates observed in the Phase 2a Study 67953964MDD2001 were less than 5% in the 2 treatment arms (4.8% in aticaprant 10 mg, and 2.4% in placebo, see Appendix 12). There was no apparent pattern of trajectories of MADRS change from baseline among participants who completed the study compared with participants who discontinued study intervention within each intervention group. Additionally, there was no specific pattern of trajectories MADRS change from baseline for each dropout reason (Appendix 12). Based on these observations, it is considered reasonable to assume missing at random (MAR) as the missingness mechanism.

MAR assumption cannot be tested vs. MNAR using observed data, however, simulation findings (Siddiqui 2009) indicate that in the presence of a mixture of the 3 missing mechanisms (missing completely at random [MCAR], MAR, missing not at random [MNAR]) with differential dropout rates between treatment groups, the MMRM approach is able to re-estimate the true treatment difference consistently with a negligible bias and control Type I error rate. Therefore, the primary analysis for this estimand will be MMRM, with sensitivity analysis using the tipping point method to stress test the efficacy findings under MNAR assumption.

## 5.3.2.1.2. Sensitivity Analysis

## Delta adjustment tipping point analysis

The sensitivity analysis for the primary Estimand – ROW will include the delta adjustment multiple imputation method which will be implemented on the MADRS total score if the results from the primary analysis show a significantly greater improvement in MADRS total score at Day 43 in aticaprant compared to placebo. This method will employ the following 3 steps:

## Step 1 – Multiple Imputation (MI)

If there are participants with a non-monotone missing data pattern, datasets with only monotone missing data patterns will be created first by imputing the intermediate missing values using methods such as the MCMC (Markov Chain Monte Carlo) method. 500 imputations will be performed to create 500 unique datasets which now have monotone missing (ie., missing data one week after the participant experienced an intercurrent event) data pattern.

Analysis assumptions: Missing at random (MAR) is assumed for intermediate missing data (i.e., missing data between non-missing observations). Monotone missing data will first be imputed by MAR-based MI regression, and the imputed scores in the experimental intervention group will be adjusted to be worse than the other participants in same group with non-missing data as discussed below. Note: Data may be monotone missing due to participant discontinuation after the ICE, or may be deemed monotone missing per the hypothetical strategy as described in Section 5.3.2 where data collected beyond one week from the occurrence of the ICE will be excluded from the primary analysis.

The imputed values will be adjusted by adding  $\delta_c$  to the imputed values for participants randomized to the control group and adding  $\delta_A$  to the imputed values for participants randomized to the experimental intervention group. Delta-adjusted fully imputed datasets will be generated for different combinations of  $\delta_c$  and  $\delta_A$  values as defined below:

•  $\delta_c = 0$  and  $\delta_A = 0$  to  $\Delta^*$  in increments of 1 (experimental group-only adjustment analysis)

Adding positive values results in higher (worse) scores.  $\Delta^*$  represents the adjustments leading to the 'tipping point', so the smallest delta adjustments values at which conclusions change from *favorable* (i.e. statistically significant: 2-sided p-value < 0.05 in favor of aticaprant) to *unfavorable* (fail to reject the null hypothesis of no intervention difference).

• Imputed values in both the experimental and the control groups will be adjusted using a range of delta values, and delta-adjusted fully imputed datasets will be generated for each combination.

These methods will be applied to all missing data under hypothetical strategy. In addition, another version of these methods will be implemented, where the delta adjustments will be applied to missing data hypothetical strategy except for those caused by discontinuation reasons due to COVID-19 (if deemed necessary), and for discontinuation reasons not related to study intervention including Lost to Follow-Up, Withdrawal by Subject or Other.

### Step 2 – Analysis

Same MMRM analysis as described for the primary efficacy analysis will be performed for each set of the adjusted fully imputed datasets.

#### Step 3 – Pooling

Rubin's methodology will be applied to the MMRM results from the 500 imputed datasets to produce final inferences.

Between-group comparisons to placebo at Day 43 (e.g. 2-sided p-values, point estimates for intervention difference) will be displayed graphically for each considered  $\delta_A$ , up to the 'tipping point' adjustment. For analysis of the imputed datasets using a range of delta-adjustments on both experimental and control groups, a tipping point two-way map will be generated.

The SAS code for the delta adjustment multiple imputation procedure is provided in Appendix 10.

#### Other sensitivity analysis

The change from baseline in MADRS total score for the primary population will be analyzed using the same MMRM model as for the primary analysis with an additional fixed effect factor for MDDANH status (MDDANH1, MDDANH2).

### 5.3.2.1.3. Other Analyses

Descriptive statistics of the observed values and the change from baseline to each time point in the double-blind and follow-up phases will be presented for MADRS total score by intervention group for FAS\_All. Change from baseline of MADRS total score will be analyzed for this analysis set using the same MMRM model as described for the primary endpoint in section along with the following additional terms in the model: ANH strata (MDDANH1, MDDANH2, MDDAH3) and age group (adult, elderly). LS mean changes from baseline (+/- SE) over time will be presented.

To assess the treatment effect in participants without anhedonia, descriptive statistics for the observed values and the change from baseline to each time point in the double-blind and follow-up phases will be presented for MADRS total score by intervention group for the MDD\_WOANH\_S and MDD WOANH MS analysis sets.

To address an FDA request to provide a supplementary analysis using a more direct measure to define moderate-to-severe anhedonia, analysis for change from baseline of MADRS total score at Day 43 for adult participants in FAS\_All will be performed in a similar manner as specified in section 5.3.2.1.1 for the sub-populations below:

• MADRS Item 8 score ( $\geq 2$ ,  $\leq 2$ )

The difference of LS mean change (95% CI) at Day 43 will be presented for each sub-population in a forest plot. Additionally, descriptive summaries of change over time in MADRS total score will be provided for the two sub-groups.

## 5.4. Secondary Endpoint(s) Analysis

The assessment of key and other secondary endpoints will be conducted on the FAS\_ANH+, which includes adult (not elderly) participants with MDD ANH+ who were randomized to aticaprant 10 mg or placebo and took at least 1 dose of study intervention, unless otherwise specified.

## 5.4.1. Key Secondary Endpoint

The key secondary efficacy endpoint is the change from baseline in DARS total score at Day 43 in FAS\_ANH+.

The same estimand (except the endpoint) and corresponding analyses as for the primary endpoint will be used for the key secondary endpoint.

## 5.4.1.1. Dimensional Anhedonia Rating Scale (DARS)

#### 5.4.1.1.1. Definition

The Dimensional Anhedonia Rating Scale (DARS) is a 17-item self-report questionnaire that was designed to assess anhedonia in MDD, and particularly to increase scale generalizability while maintaining specificity (Rizvi 2015). Respondents provide their own examples of rewarding experiences across the domains of hobbies, social activities, food/drink, and sensory experience. Participants answer a set of standardized questions about desire, motivation, effort and consummatory pleasure with a recall period of "right now" for the examples provided. Response options for each item use a 5-point Likert scale (0=not at all, 1=slightly, 2=moderately, 3=mostly, 4=very much) and responses are summed to generate the total score (range of 0 to 68) or a subscale score (range of 0 to 16 each for pastimes/hobbies, food/drink, and social activities and 0 to 20 for sensory experiences). A lower total score is indicative of greater anhedonia.

Imputation of total score is presented in Section 5.1.3.

Positive changes in DARS total score indicate improvement.

## 5.4.1.1.2. Estimand(s)

The same estimand as defined for the primary endpoint in Section 5.3.2 are defined for DARS, with the variable being the change from baseline in DARS total score at Day 43 in FAS\_ANH+.

### 5.4.1.1.3. Analysis Methods

The same analyses described for the estimand under the primary endpoint will be implemented for change from baseline in DARS total score at Day 43.

A fixed sequence testing procedure will be applied to control the family-wise error rate (FWER) at two-sided 0.05 level accounting for multiplicity due to the primary (MADRS total score) and the key secondary efficacy endpoints (DARS total score). The testing procedure will first test the primary endpoint at two-sided 0.05 level. If the hypothesis corresponding to the primary endpoint is rejected, then the key secondary endpoint will be tested at 2 sided 0.05 level; if the hypothesis corresponding to the primary endpoint is not rejected, then the testing procedure will stop.

## 5.4.1.1.4. Other Analyses

Descriptive statistics of the observed values and the change from baseline to each time point in the double-blind and follow-up phases will be presented for DARS total score by intervention group for FAS\_ANH+ and FAS\_All. Change from baseline of DARS total score based on the observed data in the double-blind phase will be analyzed for FAS\_All using the same MMRM model as described for the primary endpoint in section 5.3.2.1.1 along with the following additional terms in the model: ANH strata (MDDANH1, MDDANH2, MDDAH3) and age group (adult, elderly) LS mean changes from baseline (+/- SE) will be presented over time.

To assess the treatment effect in participants without anhedonia, descriptive statistics of the observed values and the change from baseline to each time point in the double-blind and follow-up phases will be presented for DARS total score by intervention group for MDD\_WOANH\_S and MDD WOANH MS analysis sets.

Additionally, descriptive statistics of observed values and change from baseline over time in the subscales of the DARS (hobbies/pastimes, food/drink, social activities, and sensory experiences) and proportion of participants with response at Day 43 (defined as change from baseline in DARS total score ≥ meaningful change threshold [or range of thresholds] determined by anchor-based analyses of blinded interim data) will also be provided by intervention group for FAS\_ANH+ and FAS\_All. Cumulative distribution curves for change from baseline in DARS total score by study intervention will be presented for FAS\_ANH+ and FAS\_All (Note: The meaningful change threshold, or range of thresholds, will be finalized prior to database lock).

To address an FDA request to provide a supplementary analysis using a more direct measure to define moderate-to-severe anhedonia, analysis of change from baseline of DARS total score at Day 43 for adult participants in FAS\_All will be performed in a similar manner as specified in section 5.3.2.1.1 for the following sub-populations:

• MADRS Item 8 score ( $\geq 2$ ,  $\leq 2$ )

The difference of LS mean change (95% CI) at Day 43 will be presented for each sub-population in a forest plot. Additionally, descriptive summaries of change over time in DARS total score will be provided for the two sub-groups.

## **Mediation Analysis**

A mediation analysis will be performed to examine the mediating role of change from baseline in MADRS total score at Day 43 on change from baseline in DARS total score at Day 43 provided that both endpoints demonstrate a statistically significant difference between JNJ-67953964 and placebo for FAS ANH+ under the primary estimand.

Figure 3: Meditation analysis framework



In the mediation analysis framework, natural direct effect can be conceived of as the independent treatment effect on the outcome (i.e., change in DARS total score) that is above and beyond its effect on the mediator (i.e., change in MADRS total score); controlled direct effect can be conceived of as the independent treatment effect on the outcome controlling the mediator at a fixed level; and natural indirect effect can be conceived of as a treatment effect on the outcome that is accounted for by its effect on the mediator (Figure 3).

This analysis will assess the extent to which change in DARS total score may be mediated by or independent of change in MADRS total score based on observed data (i.e., data collected at each time point without carrying forward previous values) at Day 43. The analysis will consider both change in DARS total score and change in MADRS total score as continuous variables.

Simulation-based Counterfactual Approach analysis introduced by Imai etal. (2010) obtains the natural direct effect and natural indirect effect using numerical simulations. The approach uses parametric bootstrapping to construct the point estimate and its uncertainty estimates for direct effect and indirect effect from the bootstrap sampling distribution. For each bootstrapped sample, change from baseline in DARS total score and change from baseline in MADRS total score will be analyzed. The ANCOVA analysis of change in DARS total score from baseline will include factors for intervention group (aticaprant 10 mg and placebo), country/territory, change from baseline in MADRS total score, baseline MADRS total score, treatment-by-change from baseline in MADRS total score interaction if the interaction is significant, and baseline DARS total score as a covariate. The ANCOVA analysis of change in MADRS total score will include factors for intervention group (aticaprant 10 mg and placebo) and country/territory, baseline MADRS total score and baseline DARS total score as covariates. Estimate of the controlled direct effect will be obtained by plugging in the estimated coefficient values and the mean level of change in MADRS total score into the analytic expressions.

The proposed analysis makes two important and untestable assumptions. First, the analysis is performed under the assumed causal structure shown in Figure 3, where the mediator and the outcome are measured at the same timepoint. Using cross-sectional data of this type, it is not possible to know the direction of causality (VanderWeele,2015). For example, the true causal structure may reverse the roles of mediator and outcome, where effects on anhedonia (change from baseline DARS) may mediate the effect on depressive symptoms (change from baseline MADRS). Second, to identify the natural direct and indirect effects, the analysis is performed under the standard, but untestable, assumption of sequential ignorability (Imai et al., 2010). In particular, it is assumed that the potential value of the mediator and the potential value of the outcome are independent, conditional on the treatment and any confounding variables. The impact of this second assumption will be evaluated through a sensitivity analysis as described in Tingley et al (2014).

## 5.4.2. Other Secondary Endpoint(s)

## 5.4.2.1. Response Based on MADRS Total Score

#### **5.4.2.1.1.** Definition

A participant is defined as a responder at a given time point if the percent improvement from baseline in MADRS is  $\geq 50\%$  at that time point (i.e., percent change  $\leq -50\%$ ). Participants who do not meet such criterion will be considered as non-responders. Imputation of missing response status is presented in Section 5.1.3.

#### 5.4.2.1.2. Analysis

The number and percentage of participants who achieve a response will be summarized at each time point during the double-blind phase and follow-up phase by intervention group. The summary and graph will be provided for observed and imputed data (participants with missing values will be imputed as non- responders). This analysis will be performed for FAS ANH+ analysis set.

The cumulative response rate, defined as the percentage of participants experiencing at least a given value of percent reduction from baseline to Day 43 in MADRS total score, will be presented graphically, for both observed and imputed data (participants with missing values will be imputed as non-responders).

#### 5.4.2.2. Remission Based on MADRS Total Score

#### 5.4.2.2.1. **Definition**

A participant is defined as a remitter at a given time point if the MADRS total score is  $[\le 10]$  at that time point. Participants who do not meet such criterion will be considered as non-remitters. Imputation of missing remission status is presented in Section 5.1.3.

### 5.4.2.2.2. Analysis

The number and percentage of participants who achieve remission will be summarized at each time point during the double-blind and follow-up phases by intervention group. The summary and graph will be provided for observed and imputed data (participants with missing values will be imputed as non-remitters). This analysis will be performed for FAS ANH+ analysis set.

## 5.4.2.3. Patient Health Questionnaire - 9 Item (PHQ-9)

#### 5.4.2.3.1. **Definition**



## 5.4.2.3.2. Analysis

Descriptive statistics of the observed values and the change from baseline to each time point in the double-blind and follow-up phases will be presented for PHQ-9 total score and PHQ-9 anhedonia-specific item (PHQ-9, item 1) by intervention group for FAS\_ANH+ and FAS\_All. The proportion of participants with a score >= 2 at baseline but less than 2 in the PHQ-9 anhedonia-specific item (PHQ-9, item 1) at Day 43 will be summarized for FAS\_ANH+ and FAS\_All.

The change from baseline in PHQ-9 total score over time based on the observed data in the double-blind phase will be analyzed using the same MMRM model as described for the primary endpoint with baseline PHQ-9 total score as the covariate. Difference of LS means (95% CI) will be provided at each time point.

LS mean changes from baseline (+/- SE) will be presented by over time.

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

# 5.4.2.4. PROMIS Ability to Participate in Social Roles and Activities Short Form 8a (PROMIS Social Functioning)

#### **5.4.2.4.1.** Definition



## 5.4.2.4.2. Analysis

Descriptive statistics of the observed values and the change from baseline to each time point in the double-blind and follow-up phases will be presented for the total scores of PROMIS Social Functioning Short Form 8a and the T-score by intervention group.

The change from baseline in T-score over time in the double-blind phase will be analyzed using the same MMRM model as described for the primary endpoint with baseline T-score as the covariate. Difference of LS means (95% CI) will be provided at each time point.

LS mean changes from baseline (+/- SE) for T-score will be presented graphically over time.

## 5.5. Tertiary/Exploratory Endpoint(s) Analysis

The assessment of tertiary/exploratory endpoints below will be conducted on the FAS\_ANH+ and FAS\_All separately, unless otherwise specified.

### 5.5.1.1. MADRS-6

#### 5.5.1.1.1. **Definition**



#### 5.5.1.1.2. Analysis

Descriptive statistics of the observed values and the change from baseline to each time point in the double-blind and follow-up phases will be presented for MADRS-6 total score by intervention group.

The change from baseline in MADRS-6 total score over time based on observed data in the double-blind phase will be analyzed using the same MMRM model as described for the primary endpoint with baseline MADRS-6 total score as the covariate for FAS\_ANH+. Difference of LS means (95% CI) will be provided at each time point.

LS mean changes from baseline (+/- SE) will be presented graphically over time.

# 5.5.1.2. Snaith-Hamilton Pleasure Scale (SHAPS) 5.5.1.2.1. Definition



### 5.5.1.2.2. Analysis

Descriptive statistics of the observed values and the change from baseline to each time point in the double-blind phase will be presented for SHAPS total score by intervention group.

The change from baseline of SHAPS total score over time based on the observed data in the double-blind phase will be analyzed using the same MMRM model as described for the primary endpoint with baseline SHAPS total score as a covariate for FAS\_ANH+. Difference of LS means (95% CI) will be provided at each time point.

Frequency distributions of SHAPS individual items will be provided and plotted over time in the double-blind phase for FAS ANH+.

# 5.5.1.3. Clinical Global Impression – Severity (CGI-S) 5.5.1.3.1. Definition



## 5.5.1.3.2. Analysis

Descriptive statistics of the observed values and the change from baseline will be presented at each time point in the double-blind and follow-up phases by intervention group for observed case data.

The change from baseline in CGI-S score over time based on the observed data in the double-blind phase will be analyzed using the same MMRM model as described for the primary endpoint with baseline CGI-S score as a covariate for FAS\_ANH+. Difference of LS means (95% CI) will be provided at each time point.

A frequency distribution of the CGI-S scores over time will be provided by intervention group. The frequencies of CGI-S scores will be plotted at baseline and endpoint(DB) for FAS\_ANH+.

# 5.5.1.4. Patient Global Impression of Severity (PGI-S)

#### 5.5.1.4.1. **Definition**



#### 5.5.1.4.2. Analysis

Descriptive statistics of the observed values and the change from baseline will be presented by intervention group at each time point in the double-blind and follow-up phases for observed case data for anhedonia and depression separately.

The change from baseline in PGI-S score over time based on the observed data in the double-blind phase for anhedonia and depression will be analyzed using the same MMRM model as described for the primary endpoint with baseline PGI-S score as a covariate for FAS\_ANH+. Difference of LS means (95% CI) will be provided at each time point.

LS mean changes from baseline (+/- SE) will be presented graphically over time.

A frequency distribution of the PGI-S dimension scores over time will be provided by intervention group for anhedonia and depression. The frequencies of PGI-S scores for anhedonia and depression will be plotted over time for FAS ANH+.

## 5.5.1.5. Patient Global Impression of Change (PGI-C)

#### 5.5.1.5.1. Definition



## 5.5.1.5.2. Analysis

Descriptive statistics of the observed values at endpoint in the double-blind phase will be presented by intervention group for observed case data.

An ANOVA model will be used to analyze the PGI-C score for anhedonia at endpoint(DB) between aticaprant and placebo. The model will include the PGI-C score for anhedonia at endpoint(DB) as the dependent variable, intervention group (aticaprant 10 mg and placebo) and country/territory as factors for FAS ANH+. Difference of LS means (95% CI) will be provided.

A frequency distribution of the PGI-C for anhedonia at endpoint(DB) will be provided by intervention group as well.

## 5.5.1.6. Generalized Anxiety Disorder 7-item Scale (GAD-7)

#### 5.5.1.6.1. Definition



## 5.5.1.6.2. Analysis

Descriptive statistics of the total score and change from baseline will be provided for each visit for observed data.

An ANCOVA model will be used to analyze the change from baseline in GAD-7 total score at endpoint(DB) between aticarprant and placebo for FAS\_ANH+. The model will include the change from baseline at endpoint(DB) for GAD-7 total score as the dependent variable, intervention group (aticaprant 10 mg and placebo) and country/territory as factors, and baseline GAD-7 total score as a covariate. Difference of LS means (95% CI) will be provided.

# 5.5.1.7. Quality of Life in Depression Scale (QLDS) 5.5.1.7.1. Definition



## 5.5.1.7.2. Analysis

Descriptive statistics of the total score and change from baseline will be provided for observed data.

# 5.5.1.8. European Quality of Life (EuroQol) Group, 5 Dimension, 5-Level questionnaire (EQ-5D-5L)

#### **5.5.1.8.1. Definition**


## 5.5.1.8.2. Analysis

Descriptive statistics of the observed values and the change from baseline to each time point in the double-blind and follow-up phases will be presented by intervention group for weighted EQ-5D health status index, the EQ-VAS, and the sum score.

Individual dimension responses will also be summarized at each visit with frequency counts and percentage of participants by intervention group. Proportion of participants with dimension scores of 2-5 (indicating any problem) will be plotted for each dimension at baseline and endpoint(DB) for FAS ANH+.

## 5.5.2. Subgroup Analyses

For the subgroups listed in Section 5.7.3, subgroup analyses using MMRM will be performed for the change in MADRS total score at Day 43 for FAS\_ANH+ under the primary estimand - ROW. The fixed terms in the model will be intervention group, country/territory, time, subgroup, time-by-intervention interaction, intervention-by-subgroup interaction, and time-by-intervention-by-subgroup interaction, and baseline MADRS total score as a covariate. Point estimates of the treatment differences and 2-sided 95% CI will be estimated using the appropriate contrasts. Country/territory will not be included in the model if the subgroup of interest is Region.

The analysis results (difference of LS means and 95% CI) of the different subgroups will be displayed in a forest plot.

Similar analyses will be performed for the change in DARS total score at Day 43 and the results will be displayed in a forest plot.

### 5.6. Safety Analyses

All safety analyses will be based on safety analysis set based on randomized intervention, unless otherwise specified.

Safety analysis will be conducted separately for the DB and follow-up phases.

CONFIDENTIAL – FOIA Exemptions Apply in U.S.

For all continuous safety variables, descriptive statistics by intervention group will include the N, mean, standard deviation, median, minimum, and maximum. Categorical variables will be summarized by intervention group using frequency counts and percentages.

## 5.6.1. Extent of Exposure

The number and percentage of participants who receive study intervention will be summarized.

Descriptive statistics for duration of study intervention and of the current antidepressant (N, mean, SD, median, and range (minimum, maximum)) will be summarized.

Duration of study intervention will be summarized in the following categories: <=7 days, 8-14 days, 15-21 days, 22-28 days, 29-35 days, 36-42 days, >42 days.

Study intervention duration is defined as (date of last dose of study intervention – date of first dose of study intervention) +1. Total number of dosing days is defined as the total number of days the study intervention was administered to the participant (excluding days off study intervention).

Current antidepressant duration is defined as (minimum of end of double-blind study intervention and end of antidepressant use – maximum of start of double-blind study intervention and start of antidepressant use)+1.

The summaries will be provided for FAS\_ANH+, MDD\_WOANH\_S, MDD\_WOANH\_MS and safety analysis set.

#### **5.6.1.1.** Compliance

Compliance will be summarized descriptively for each study intervention and the current antidepressant.

The percent compliance will be categorized (<60%, 60-<80%, 80-<100%, 100%) and the number and percentage of participants in each category will be summarized for study intervention and for the current antidepressant.

Compliance will be calculated for the study intervention as:

Compliance (%) = (number of days when participant took the expected number of large tablets) / (duration of study intervention)  $\times 100\%$ 

Compliance will be calculated for the current antidepressant as:

Compliance (%) = (number of days actually dosed with the current antidepressant while on study intervention) / (duration of study intervention)  $\times 100\%$ 

The summaries will be provided for FAS\_ANH+, MDD\_WOANH\_S, MDD\_WOANH\_MS and safety analysis sets.

#### 5.6.2. Adverse Events

The verbatim terms used in the CRF by investigators to identify adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). Any AE occurring at or after the initial administration of study intervention through the end of DB phase is considered to be treatment emergent. If the event occurs on the day of the initial administration of study intervention (and action taken is not entered as 'Not Applicable' in the database), then the event will be considered as treatment emergent. If the event date is recorded as partial or completely missing, then the event will be considered to be treatment emergent unless it is known to be prior to the first administration of study intervention based on partial onset date or resolution date. All reported adverse events will be included in the analysis. For each adverse event, the number and percentage of participants who experience at least 1 occurrence of the given event will be summarized by intervention group.

Assignment of adverse events to the appropriate phase will be made based on the following rules:

#### **Double-blind treatment phase:**

AEs during the DB phase will satisfy the condition: DB phase start date  $\leq$  AE onset date  $\leq$  DB phase end date.

#### Follow-up phase:

AEs that are assigned to the follow-up phase will not be considered as treatment-emergent. AEs during the follow-up phase will satisfy the condition: follow-up phase start date  $\leq$  AE onset date  $\leq$  follow-up phase end date.

Summary tables will be provided for:

- AEs (all AEs, and AEs with incidence of at least 5% in any treatment group)
- Serious AEs (SAEs)
- AEs leading to discontinuation of study intervention (DB treatment phase only)
- AEs by severity
- AEs by relationship to study intervention
- Severe AEs
- AEs of special interest



- AEs of clinical interest
  - o system organ class AEs
  - Suicide/Self-injury (First Sub SMQ)
  - o AEs suggestive of abuse potential (Appendix 11)

In addition to the summary tables, listings will be provided for participants who:

- Died
- Had SAEs
- Had AEs leading to discontinuation of study intervention
- Had AEs of special interest

- Special interest AEs include CCI
- · Had AEs of clinical interest
  - o system organ class AEs
  - Suicide/Self-injury (First Sub SMQ)
  - o AEs suggestive of abuse potential

In addition, for each AESI, the number of days of dosing prior to onset, duration of the event, frequency distribution of the number of occurrences, and number of participants who were treated with concomitant medications will be summarized.

#### 5.6.3. Additional Safety Assessments

#### 5.6.3.1. Clinical Laboratory Tests

Descriptive statistics will be presented for all chemistry, hematology, and urinalysis laboratory tests at scheduled time points in the double-blind phase.

Change from baseline to all post-baseline visits in the double-blind phase will be summarized for chemistry, hematology, and urinalysis tests and displayed by study intervention group.

Clinical laboratory test values collected in the double-blind phase will be considered "treatment-emergent markedly abnormal" (TEMA) using the criteria defined by the sponsor listed in Appendix 8.

- If the postbaseline value is above the upper limit of the markedly abnormal criteria and the baseline value is below the upper limit, then the postbaseline marked abnormality will be considered TE. The same applies to the postbaseline value being below the lower limit of the markedly abnormal criteria with the baseline value being above the lower limit of the markedly abnormal criteria.
- If the baseline value is missing, a postbaseline marked abnormality will always be considered as TF.

The number and percentage of participants with treatment-emergent markedly abnormal values will be presented by study intervention group. It will be conducted for all participants and separately for the participants who experience TEAEs.

Incidence of participants with ALT values  $\geq$  3\*upper normal limit (ULN), AST values  $\geq$  3\*ULN, total bilirubin values  $\geq$  2\*ULN (or at least doubling of direct bilirubin in known Gilbert's syndrome),, and international normalized ratio (INR) > 1.5 (if measured) will be presented for the double-blind phase. Additionally, incidence of hepatic toxicity (Hy's Law) defined as ALT or AST values  $\geq$  3\*ULN AND alkaline phosphatase < 2\*ULN AND (total bilirubin values  $\geq$  2\*ULN OR international normalized ratio (INR) > 1.5, if measured) in the double-blind phase will be presented. Participants with baseline (DB) values meeting these criteria will not be considered as having treatment-emergent hepatic toxicity.

A listing of participants with markedly abnormal laboratory values will be provided for the double-blind phase. A listing of participants with ALT  $\geq$  3\* ULN or AST values  $\geq$  3\*ULN) and participants with hepatic toxicity (suspected Hy's Law cases) in the double-blind phase will be provided.

## 5.6.3.2. Vital Signs and Physical Examination Findings

Continuous vital sign parameters including temperature, weight, pulse, blood pressure (systolic and diastolic), and Body Mass Index (BMI) will be summarized at each assessment time point. Body Mass Index will be calculated as weight (kg)/(height (m))<sup>2</sup>, at each time point that body weight is measured. The height measurement collected at screening will be used in the calculation. Change from the baseline will be summarized over time. Descriptive statistics (mean, standard deviation, median, minimum and maximum) will be presented.

Abnormality criteria (based on criteria defined below) will be applied to postbaseline values in the double-blind phase.

Postbaseline values will be considered treatment-emergent if they meet both value and change criteria in the table below.

For criteria that do not include an increase or decrease from baseline:

- Treatment-emergent will be concluded if the postbaseline value is above the upper limit and the baseline value is below the upper limit (eg, Normal or Low). The same applies to the postbaseline value being below the lower limit with the baseline value being above the lower limit (eg, Normal or High).
- If the baseline value is missing, a postbaseline abnormality will always be considered as TE.

Incidence of treatment-emergent clinically important vital signs during intervention, as defined in Table 4, will be summarized for participants who had a baseline assessment and at least 1 postbaseline assessment for that vital sign during the DB phase. A listing of participants with treatment-emergent clinically important abnormalities in vital signs during the DB phase will be presented, along with a listing of clinical important vital sign measurements.

**Table 4: Clinically Important Abnormalities in Vital Signs** 

| Vital Sign | <b>Abnormal Category</b> | Criteria |
|---|---|---|
| Pulse | Abnormally high | ≥100 bpm and with ≥15 bpm increase from baseline |
| | Abnormally low | ≤50 bpm and with ≥15 bpm decrease from baseline |
| Systolic blood pressure | Abnormally high | ≥180 mm Hg and with ≥20 mm Hg increase from baseline |
| | Abnormally low | ≤90 mm Hg and with ≥20 mm Hg decrease from baseline |
| Diastolic blood pressure | Abnormally high | ≥105 mm Hg and with ≥15 mm Hg increase from baseline |
| | Abnormally low | ≤50 mm Hg and with ≥15 mm Hg decrease from baseline |
| Temperature | Abnormally high | >37.5°C |
| | Abnormally low | <35.5°C |
| Weight | Abnormally high | increase ≥7% from baseline |
| | Abnormally low | decrease ≥7% from baseline |

## 5.6.3.3. Electrocardiogram

The ECG parameters that will be analyzed are heart rate, PR interval, QRS interval, QT interval, and corrected QT (QTc) interval using the following correction methods: Bazett's formula (QTcB), Fridericia's formula (QTcF).

Bazett's formula: QTcB (msec) = QT (msec) /  $(RR (msec)/1000)^{1/2}$ ; if RR is missing, use QT (msec) \*  $(HR(bpm)/60)^{1/2}$ ;

Fridericia's formula: QTcF (msec) = QT (msec) / (RR (msec)/1000)<sup>1/3</sup>; if RR is missing, use QT (msec) \*  $(HR(bpm)/60)^{1/3}$ ;

Baseline is the most recent assessment prior to the first dose, or average of the most recent assessments prior to the first dose if multiple assessments are done on the same day.

The number and percentage of participants with QTc interval will be summarized at each time point in the double-blind phase. The number and percentage of participants with QTc interval increases from baseline to the maximum postbaseline value and each post dose time point will be summarized for double-blind phase. Refer to the following Table 5 for summary categories.

| Parameter | Classification | Criteria |
|---|---|---|
| QTc change from baseline | No concern | ≤30 |
| | Concern | >30 - 60 |
| | Clear concern | > 60 |
| QTc value | Normal | ≤450 for male,<br>≤470 for female |
| | > 450 – 480 for male,<br>> 470 – 480 for female | >450 to ≤480 for male,<br>>470 to ≤480 for female |
| | > 480 - 500 | >480 - ≤500 |
| | > 500 | > 500 |

Table 5: Criteria for Abnormal QTc Values and Changes From Baseline

Shift table will be provided from baseline to maximum post baseline QTc interval for the double-blind phase.

Descriptive statistics of ECG parameters and change from baseline will be summarized at each scheduled time point for double-blind and follow-up phases.

Abnormality criteria (based on criteria defined in Table 6 below) will be applied to baseline and postbaseline values in the double-blind phase.

Postbaseline abnormalities will be compared with their corresponding baseline result:

- Treatment-emergent will be concluded if the postbaseline value is above the upper limit and the baseline value is below the upper limit (eg, Normal or Low). The same applies to the postbaseline value being below the lower limit with the baseline value being above the lower limit (eg, Normal or High).
- If the baseline value is missing, a postbaseline abnormality will always be considered as treatment-emergent.

The number and percentage of participants with treatment-emergent ECG values outside predefined limits will be presented by study intervention over time for the double-blind phase:

**Table 6: Abnormal Limits for ECG Parameters** 

| | Outside | Outside of normal limit if |
|---------------------|----------------|----------------------------|
| ECG Parameter | Abnormally low | Abnormally high |
| Heart Rate (bpm) | ≤ 50 bpm | ≥100 bpm |
| PR interval (msec) | ≤ 120 msec | ≥ 200 msec |
| QRS interval (msec) | ≤ 60 msec | ≥120 msec |
| QT interval (msec) | ≤ 200 msec | ≥500 msec |
| RR interval (msec) | < 600 msec | > 1200 msec |

The interpretation of the ECGs as determined by a central reader will be displayed by the number and percentage of participants meeting the normality criteria. The interpretation will be summarized over time.

Listings of ECG abnormalities (see Table 6) and abnormal QTc values in the double-blind phase will also be provided.

## 5.6.3.4. Other Safety Parameters

#### 5.6.3.4.1. Columbia Suicide Severity Rating Scale (C-SSRS)





#### 5.6.3.4.3. Physician Withdrawal Checklist 20-item (PWC-20)



#### 5.7. Other Analyses

#### 5.7.1. Pharmacokinetics

PK analyses will be performed on the safety analysis set.

Descriptive statistics (N, mean, SD, median, range, CV (%) and IQ range) will be used to summarize plasma concentrations at each sampling time point and for each PK parameter of Active Study Intervention.

#### 5.7.2. Biomarkers

Analysis of biomarker data will be discussed in a separate SAP.

#### 5.7.3. Definition of Subgroups

Subgroup analyses of the primary and key secondary endpoints will be performed for the FAS\_ANH+ analysis sets for the following subgroups:

- Sex (male, female, unknown, undifferentiated)
- Race (Black or African American, White, Other, Not Reported)
- Ethnicity (Hispanic or Latino, not Hispanic or Latino, Not Reported, Unknown)
- Country/territory
- Region (south America, north America, Europe, other)
- Age Group (18-44 years, 45-64 years)
- BMI (underweight  $<18.5 \text{ kg/m}^2$ , normal 18.5- $<25 \text{ kg/m}^2$ , overweight 25- $<30 \text{ kg/m}^2$ , obese  $>=30 \text{ kg/m}^2$ )
- Number of major depressive episodes (1, 2-5, 6-10, >10)
- Curent antidepressant type (SSRI, SNRI)
- Baseline MADRS (≤/> median)
- Baseline DARS (≤/>median)

- Benzodiazepine (Yes, No)
- SCID-CT With melancholic features (Yes, No)
- SCID-CT With anxious distress (Yes, No)

## 5.8. Interim Analyses

A blinded interim analysis will be performed to evaluate the measurement properties of the DARS, and to determine meaningful change threshold (MCT) (or range of thresholds) in the DARS total score using anchor-based approaches along with distribution-based analyses. The interim analysis will be conducted when approximately 200 adult MDD participants, regardless of anhedonia status, have completed the DB Treatment Phase of the study. Details of the analysis will be described in a separate analysis plan.

## 5.8.1. Independent Data Monitoring Committee (IDMC)

An Independent Data Monitoring Committee (IDMC) will be commissioned to periodically review safety data for this study. Details about the membership of the IDMC and its roles and responsibilities are discussed in a separate IDMC charter.

#### 6. SUPPORTING DOCUMENTATION

## 6.1. Appendix 1 List of Abbreviations

| AESI Adverse event() of special interest ALT Alanine aminotransferase ANCOVA Analysis of covariance ASEX Arzona Sexual Maturity Scale AST Aspartate aminotransferase BMI Body mass index C-SSRS Columbia suicide severity rating scale CGSSRS Columbia suicide severity rating scale CGI-S Clinical global impression-severity CI Confidence interval CIR Copy increment from reference CR Copy increment from reference CR Copy effectence CRF Case report form CV Coefficient of variation DARS Dimensional anhedomia rating scale DB Double-blind DB Data Presentation Specifications DSM-5 Diagnostic and statistical manual of mental disorders, 5th edition ECG Electrocardiogram ECG | | Statistical Analysis Plan 0/955904WIDD5002 |
|---|---|---|
| ALT Alamine aminotransferase ANCOVA Analysis of covariance ASEX Arizona Sexual Maturity Scale AST Aspartate aminotransferase AST Aspartate aminotransferase AST Aspartate aminotransferase AST Aspartate aminotransferase BMI Body mass index C-SSRS Columbia suicide severity rating scale CGI-SSRS Columbia suicide severity rating scale CGI-S Clinical global impression-severity CI Confidence interval CIR Copy increment from reference CR Copy increment from reference CR Copy reference CRF Case report from CV Coefficient of variation DARS Dimensional anhedonia rating scale DB Double-blind DPS Data Presentation Specifications DSM-5 Diagnostic and statistical manual of mental disorders, 5th edition ECG Electrocardiogram ECG Electrocardiogram EQ-5D-5L European quality of life, 5-dimension, 5-level EQ-VAS European quality of life, 5-dimension, 5-level EQ-VAS European quality of life visual analog scale EU European union FAS ANI Full analysis set (AII) FAS ANH Full Analysis set (AII) FAS ANH Full Analysis set (AII) FAS ANH Full Analysis set (AII) FU Follow-up FWER Familywise error rate GAD-7 Generalized auxiety disorder 7-item scale GI Gastrointestinal HSI Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile ILS Least squares MADRS Montgomery-asherg depression rating scale MADR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD ANH MDD with moderate-to-severe anhedonia MDD ANH MDD with moderate-to-severe anhedonia MDD WOANH S MDD without anhedonia SI MCD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia SI MCD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedoni | AE | Adverse event |
| ANCOVA Analysis of covariance ASEX Arizona Sexual Maturity Scale AST Aspartate aminotransferase ATC Anatomic and therapeutic class BMI Body mass index C-SSRS Columbia suicide severity rating scale C-SSRS Colimical global impression-severity CI CI Confidence interval CIR Copy increment from reference CRR Copy reference CRR Copy reference CRF Case report form CV Coefficient of variation DARS Dimensional anhedonia rating scale DB Double-blind DFS Data Presentation Specifications DSM-5 Diagnostic and statistical manual of mental disorders, 5th edition ECG EIectrocardiogram ECG EIectrocardiogram ECG EQ-VAS European quality of life-yisual analog scale EU European union FAS AII Full analysis set (AII) FAS ANH+ Full Analysis Set (ANH+) FU Follow-up FWER Familywise error rate GAD-7 Generalized anxiety disorder 7-item scale GI GI Gastoriottestinal HSI Health status index IICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ International Conference on Harmonisation IDMC Markov chain monte carlo MCM MAR Missing at random MCMC Markov chain monte carlo MCMC Markov chain monte | AESI | Adverse event(s) of special interest |
| ASEX Airona Sexual Maturity Scale AST Aspartate aminotransferase ATC Anatomic and therapeutic class BMI Body mass index CSSRS Columbia suicide severity rating scale CGI-S Clinical global impression-severity CI Confidence interval CIR Copy increment from reference CR Copy reference | ALT | Alanine aminotransferase |
| AST Aspartate aminotransferase ATC Anatomic and therapeutic class BMI Body mass index C-SSRS Columbia suicide severity rating scale CGG-S Clinical global impression-severity CI Confidence interval CIR Copy increment from reference CR Copy reference CP Physician Global mpression-Change CDL South of the reference CR Copy reference CR Co | ANCOVA | Analysis of covariance |
| ATC Anatomic and therapeutic class BMI Body mass index C-SSRS Columbia suicide severity rating scale CGF-S Climical global impression-severity CI Confidence interval CIR Copy increment from reference CR Copy reference CRF Case report form CV Coefficient of variation DARS Dimensional anhedomia rating scale DB Double-blind DPS Data Presentation Specifications DSM-5 Diagnostic and statistical manual of mental disorders, 5th edition ECG Electrocardiogram EQ-SD-5L European quality of life, 5-dimension, 5-level EQ-VAS European quality of life, 5-dimension, 5-level EU European union FAS All Full analysis set (All) FAS ANH+ Full Analysis Set (ANH+) FU Follow-up FWER Familywise error rate GAD-7 Generalized anxiety disorder 7-item scale GI Gastrointestinal HSI Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IL EL Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MDD ANH- MDD without anhedonia MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH MS MDD without anhedonia MMRM Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs Non-steroidal anti-inflammatory drugs Non-steroidal anti-inflammatory drugs Non-steroidal anti-inflammatory drugs Non-Steroidal anti-inflammatory dru | ASEX | Arizona Sexual Maturity Scale |
| ATC Anatomic and therapeutic class BMI Body mass index C-SSRS Columbia suicide severity rating scale CGF-S Climical global impression-severity CI Confidence interval CIR Copy increment from reference CR Copy reference CRF Case report form CV Coefficient of variation DARS Dimensional anhedomia rating scale DB Double-blind DPS Data Presentation Specifications DSM-5 Diagnostic and statistical manual of mental disorders, 5th edition ECG Electrocardiogram EQ-SD-5L European quality of life, 5-dimension, 5-level EQ-VAS European quality of life, 5-dimension, 5-level EU European union FAS All Full analysis set (All) FAS ANH+ Full Analysis Set (ANH+) FU Follow-up FWER Familywise error rate GAD-7 Generalized anxiety disorder 7-item scale GI Gastrointestinal HSI Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IL EL Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MDD ANH- MDD without anhedonia MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH MS MDD without anhedonia MMRM Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs Non-steroidal anti-inflammatory drugs Non-steroidal anti-inflammatory drugs Non-steroidal anti-inflammatory drugs Non-Steroidal anti-inflammatory dru | AST | Aspartate aminotransferase |
| BMI Body mass index C-SSRS Columbia suicide severity rating scale CGI-S Clinical global impression-severity CI Confidence interval CIR Copy increment from reference CR Copy increment from reference CRF Case report form CV Coefficient of variation DARS Dimensional anhedonia rating scale DB Double-blind DPS Data Presentation Specifications DSM-5 Diagnostic and statistical manual of mental disorders. 5th edition ECG Electrocardiogram ECG Electrocardiogram ECG Electrocardiogram EQ-SD-51. European quality of life, 5-dimension, 5-level EQ-VAS European quality of life, 5-dimension, 5-level EQ-VAS European quality of life, 5-dimension, 5-level EU European union FAS All Full analysis set (AII) FAS ANH+ Full Analysis Set (ANH+) FU Follow-up FWER Familywise error rate GAD-7 Generalized anxiety disorder 7-item scale GI Gastrointestinal HSI Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Montgomery-asberg depression rating scale MARR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD ANH- MDD without moderate-to-severe anhedonia MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH S MDD without anhedonia MNAR Missing not at random MNAR Missing not at random MNAR Missing not at random NSAIDS Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGG-C Physician Global Impression-Change PG-S Physician Global Impression-Change PG-S Physician Global Impression-Severity PHO-O Paleint Health Questionnaire-9 Hem PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS | | • |
| C-SSRS Columbia suicide severity rating scale CGI-S Clinical global impression-severity CI COnfidence interval CIR Copy increment from reference CR CR Copy reference CRF Case report form CV Coefficient of variation DARS Dimensional anhedonia rating scale DB Double-blind DPS Data Presentation Specifications DSM-5 Diagnostic and statistical manual of mental disorders, 5th edition ECG Electrocardiogram EQ-SD-51 European quality of life, 5-dimension, 5-level EQ-SD-51 European quality of life-visual analog scale EU European quality of life-visual analog scale EU European quality of life-visual analog scale EU European quality of life-visual analog scale EU European quality of life-visual analog scale FAS All Full analysis set (All) FAS ANH+ Full Analysis set (All) FAS ANH+ Full Analysis set (All) FAS Collow-up FWER Familywise error rate GAD-7 Generalized anxiety disorder 7-item scale GI Gastrointestinal HSI Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD Major depressive disorder MDD ANH+ MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH MS MDD without anhedonia MNAR Missing not at random NSAIDS Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 tem PK Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 tem PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items | | • |
| CGI-S CInical global impression-severity CI COnfidence interval CIR Copy increment from reference CR COpy reference CR Copy reference Cappending Copy reference Copy reference Cappending Copy reference | | ř |
| CI CIR Copy increment from reference CR CR Copy reference CRF Case report form CV Coefficient of variation DARS Dimensional anhedonia rating scale DB Double-blind DPS Data Presentation Specifications DSM-5 Diagnostic and statistical manual of mental disorders, 5th edition ECG EICG Electrocardiogram EQ-5D-51. European quality of life, 5-dimension, 5-level EQ-VAS European quality of life-visual analog scale EU European quality of life-visual analog scale EU European quality of life-visual analog scale EU European quality of life-visual manual of mental disorders, 5th edition FAS All Full analysis set (All) FAS ANH+ Full Analysis Set (ANH+) FU FOU FOIlow-up FWER Familywise error rate GAD-7 Generalized anxiety disorder 7-item scale GI Gastrointestinal HSI Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD Major depressive disorder MDD ANH- MDD without anhedonia MDD WANH M MDD without moderate-to-severe anhedonia MDD WANH M MDD without moderate-to-severe anhedonia MDD WANH M MDD without anhedonia MDD WANH M MDD without anhedonia MDD WANH M MDD without anhedonia MDD WANH M MDD without anhedonia MDD WANH M MDD without anhedonia MDD WANH M MSmign got at random MNAR Missing nat random MNAR Missing nat random NSAIDS Non-steroidal anti-inflammatory drugs NSAIDS Non-steroidal anti-inflammatory drugs NSAIDS Non-steroidal anti-inflammatory drugs NSAIDS Non-steroidal anti-inflammatory drugs NSAIDS Non-steroidal anti-inflammatory drugs NSAIDS Physician Global Impression-Severity PHQ-9 Patient Health Questionaniar-9 ftem PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS | | |
| CIR Copy increment from reference CR Copy reference CRF Case report form CV Coefficient of variation DARS Dimensional anhedonia rating scale DB Double-blind DPS Data Presentation Specifications DSM-5 Diagnostic and statistical manual of mental disorders, 5th edition ECG Electrocardiogram EQ-515-1L European quality of life, 5-dimension, 5-level EQ-VAS European quality of life-visual analog scale EU European quality of life-visual analog scale EU European union FAS All Full analysis set (All) FAS ANH+ Full Analysis set (ANH+) FU Follow-up FWER Familywise error rate GAD-7 Generalized anxiety disorder 7-item scale GI Gastrointestinal HSI Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD MAH MDD with underate-to-severe anhedonia MDD MOANH MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH MS MDD without anhedonia MDD | | |
| CR CRF Case report form CV Coefficient of variation DARS Dimensional anhedonia rating scale DB Double-blind DPS Data Presentation Specifications DSM-5 Diagnostic and statistical manual of mental disorders, 5th edition ECG Electrocardiogram EQ-5D-5L European quality of life, 5-dimension, 5-level EQ-VAS European quality of life-visual analog scale EU European union FAS All Full analysis set (All) FAS ANH+ Full Analysis set (All) FVAS European quality of life-visual analog scale EU European union FAS All Full analysis set (All) FVAS European quality of life-visual analog scale EU European union FAS ANH+ Full Analysis set (All) FVAS European quality of life-visual analog scale EU European union FAS ANH+ Full Analysis set (All) FVAS European quality of life-visual analog scale EU European union FAS ANH+ Full Analysis set (All) FVAS EVAS European quality of life-visual analog scale EVAS European quality of life-visual analog scale EVAS EUROPEAN EVAS EUROPEAN EVAS EUROPEAN EVAS EUROPEAN EVAS EVAS EVAS EUROPEAN EVAS | | |
| CRF CV Coefficient of variation DARS Dimensional anhedonia rating scale DB Double-blind DPS Data Presentation Specifications DSM-5 Diagnostic and statistical manual of mental disorders, 5th edition ECG Electrocardiogram EQ-51D-51 European quality of life, 5-dimension, 5-level EQ-VAS European quality of life, 5-dimension, 5-level EU European quality of life-visual analog scale EU European union FAS All Full analysis set (All) FAS ANH+ Full Analysis set (ANH+) FU FOI FOIlow-up FWER Familywise error rate GAD-7 Generalized anxiety disorder 7-item scale GI Gastrointestinal HSI Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD MSH MDD MANH- MDD with moderate-to-severe anhedonia MDD ANH- MDD without anhedonia MDD MOANH S MDD without anhedonia MDD | | |
| CV Coefficient of variation DARS Dimensional anhedonia rating scale DB Double-blind DPS Data Presentation Specifications DSM-5 Diagnostic and statistical manual of mental disorders, 5th edition ECG Electrocardiogram EQ-5D-5L European quality of life, 5-dimension, 5-level EQ-VAS European quality of life, 5-dimension, 5-level EU European quality of life-visual analog scale EU European quality of life life-visual analog scale | | |
| DARS Dimensional anhedonia rating scale DB Double-blind DPS Data Presentation Specifications DSM-5 Diagnostic and statistical manual of mental disorders, 5th edition ECG Electrocardiogram EQ-5D-5L European quality of life, 5-dimension, 5-level EQ-VAS European quality of life, 5-dimension, 5-level EQ-VAS European quality of life, 5-dimension, 5-level EU European union FAS AII Full analysis set (AII) FAS ANH+ Full Analysis set (ANH+) FU Follow-up FWER Pamilywise error rate GAD-7 Generalized anxiety disorder 7-item scale GI Gastrointestinal Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Monigomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD MARH MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH MS MDD without anhedonia MI Multiple imputation MMRM Miscd model for repeated measures MNAR Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) Quality of life in depression scale | | |
| DB Double-blind DPS Data Presentation Specifications DSM-5 Diagnostic and statistical manual of mental disorders, 5th edition ECG Electrocardiogram EQ-5D-5L European quality of life, 5-dimension, 5-level EQ-VAS European quality of life, visual analog scale EU European union FAS All Full analysis set (All) FAS ANH+ Full Analysis Set (ANH+) FU Follow-up FWER Familywise error rate GAD-7 Generalized anxiety disorder 7-item scale GI Gastrointestinal HSI Health status index ICH International Conference on Harmonisation DMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Monigomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD Major depressive disorder MDD ANH+ MDD with moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH MI Mixed model for repeated measures MNAR Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs Non-ster | | |
| DPS Data Presentation Specifications DSM-5 Diagnostic and statistical manual of mental disorders, 5th edition ECG Electrocardiogram EQ-5D-5L European quality of life, 5-dimension, 5-level EQ-VAS European quality of life-visual analog scale EU European quality of life-visual analog scale EU European quality of life-visual analog scale EU European quality of life-visual analog scale EU Full analysis set (All) FAS All Full analysis set (ANH+) FU Follow-up FWER Familywise error rate GAD-7 Generalized anxiety disorder 7-item scale GI Gastrointestinal HSI Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile IS Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD MAH+ MDD with moderate-to-severe anhedonia MDD ANH+ MDD with moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH MS MDD without anhedonia MGMRM Mixed model for repeated measures MNAR Missing not at random NSAIDS Non-steroical anti-imflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | |
| DSM-5 Diagnostic and statistical manual of mental disorders, 5th edition ECG Electrocardiogram EQ-5D-5L European quality of life, 5-dimension, 5-level EQ-VAS European quality of life-visual analog scale EU European quality of life-visual analog scale EU European union FAS All Full analysis set (All) FAS ANH+ Full Analysis Set (ANH+) FU Follow-up FWER Familywise error rate GAD-7 Generalized anxiety disorder 7-item scale GI Gastrointestinal HSI Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD ANH- MDD with moderate-to-severe anhedonia MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without moderate-to-severe anhedonia MMRM Missing not at random MMRM Missing not at random MNAR Missing not at random MNAR Missing not at random NNAR Missing not at random NNAR Missing not at random NNAR Missing not at random NNAR Missing not at random NNAR Missing not at random NSAIDS Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | |
| ECG Electrocardiogram EQ-5D-5L European quality of life, 5-dimension, 5-level EQ-VAS European quality of life-visual analog scale EU European union FAS All Full analysis set (All) FAS ANH+ Full Analysis Set (ANH+) FU Follow-up FWER Familywise error rate GAD-7 Generalized anxiety disorder 7-item scale GI Gastrointestinal HSI Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD Major depressive disorder MDD ANH+ MDD with moderate-to-severe anhedonia MDD ANH- MDD without anhedonia MDD WOANH S MDD without anhedonia MEMD Medical Dictionary for Regulatory Activities MI Multiple imputation MNAR Missing not a random MNAR Missing not a random MNAR Missing not at a random MNAR Missing not at a random MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MRM Missing not at random MNAR Missing not at random NNAR Missing not at random NNAR Missing not at random NNAR Missing not at random NNAR Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-C Physician Global Impression-Change PGI-C Physician Global Impression-Change PK Pharmacokinetic(s) PMC-20 Physician Withdrawal Checklist 20-items QLDS | | |
| EQ-5D-5L European quality of life, 5-dimension, 5-level EQ-VAS European quality of life-visual analog scale EU European union FAS All Full analysis set (All) FAS ANH Full Analysis Set (ANH+) FU Follow-up FWER Familywise error rate GAD-7 Generalized anxiety disorder 7-item scale GI Gastrointestinal HSI Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD ANH+ MDD with moderate-to-severe anhedonia MDD ANH+ MDD without anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH MS MDD without anhedonia MDD Wollow Mealon of Regulatory Activities MI Multiple imputation MNAR Missing not at random MNAR Missing not at random MNAR Missing not at random MNAR Medical Dictionary for Regulatory Activities MI Multiple imputation MNRM Mixed model for repeated measures MNAR Missing not at random NSAIDS Non-steroidal anti-inflammatory drugs Non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | , |
| EQ-VAS European quality of life-visual analog scale EU European union FAS All Full analysis set (All) FAS ANH+ Full Analysis Set (ANH+) FU Follow-up FWER Familywise error rate GAD-7 Generalized anxiety disorder 7-item scale GI Gastrointestinal HSI Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Monitgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD ANH+ MDD with moderate-to-severe anhedonia MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MI Multiple imputation MMRM Missing not at random MNAR Missing not at random MNAR Medical Dictionary for Regulatory Activities MI Multiple imputation MNAR Missing not at random NSAIDS Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-C Physician Global Impression-Change PGI-C Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) Quality of life in depression scale | | |
| EU European union FAS All Full analysis set (All) FAS ANH+ Full Analysis Set (ANH+) FU Follow-up FWER Familywise error rate GAD-7 Generalized anxiety disorder 7-item scale GI Gastrointestinal HSI Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Montgomery-asberg depression rating scale MARR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD Major depressive disorder MDD ANH+ MDD with moderate-to-severe anhedonia MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH S MDD without anhedonia MED MOANH Medical Dictionary for Regulatory Activities MI Multiple imputation MNAR Missing not at random NNAR Missing not at random NNAR Missing not at random NNAR Missing not at random NSAIDS Non-steroidal anti-inflammatory drugs Non-PAP Non primary analysis population PGI-C Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PUC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | |
| FAS All Full analysis set (All) FAS ANH+ Full Analysis Set (ANH+) FU Follow-up FWER Familywise error rate GAD-7 Generalized anxiety disorder 7-item scale GI Gastrointestinal Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD Major depressive disorder MDD ANH+ MDD with moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH S MDD without anhedonia MEDRA Medical Dictionary for Regulatory Activities MI Multiple imputation MNRRM Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PKC Physician Global Impression-Change PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PUC-20 Physician Withdrawal Checklist 20-items VALUE PAIL AND TIME TO THE | | 1 1 7 |
| FAS_ANH+ Full Analysis Set (ANH+) FU Follow-up FWER Familywise error rate GAD-7 Generalized anxiety disorder 7-item scale GI Gastrointestinal HSI Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD ANH+ MDD with moderate-to-severe anhedonia MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MOD without anhedonia MDRA Medical Dictionary for Regulatory Activities MI Multiple imputation MMRM Mixed model for repeated measures MNAR Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) QLDS Quality of life in depression scale | | • |
| FUER Familywise error rate GAD-7 Generalized anxiety disorder 7-item scale GI Gastrointestinal HSI Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD Major depressive disorder MDD ANH+ MDD with moderate-to-severe anhedonia MDD ANH+ MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH S MDD without anhedonia MEDRA Medical Dictionary for Regulatory Activities MI Multiple imputation MMRM Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionmaire-9 Item PK Pharmacokinetic(s) Quality of life in depression scale | | • • • |
| FWER GAD-7 Generalized anxiety disorder 7-item scale GI Gastrointestinal HSI Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD Major depressive disorder MDD ANH+ MDD with moderate-to-severe anhedonia MDD ANH- MDD without anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MDRA Medical Dictionary for Regulatory Activities MI Multiple imputation MMRM Mixed model for repeated measures MNAR Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS QLDS Gastrointesian Harmonisation International Conference on Harmonisation International Conference on Harmonisation Ha | | , , , |
| GAD-7 Generalized anxiety disorder 7-item scale GI Gastrointestinal HSI Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD Major depressive disorder MDD ANH+ MDD with moderate-to-severe anhedonia MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH S MDD without anhedonia MMDM MedDRA Medical Dictionary for Regulatory Activities MI Multiple imputation MMRM Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | • |
| GI Gastrointestinal HSI Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD Major depressive disorder MDD ANH+ MDD with moderate-to-severe anhedonia MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MOD without anhedonia MCI MCT MARCH MARCH MISSING MARCH MISSING Non-steroidal anti-inflammatory drugs NON-SEROIDAL AND MISSING NON-steroidal anti-inflammatory drugs NON-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | |
| HSI Health status index ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD Major depressive disorder MDD ANH+ MDD with moderate-to-severe anhedonia MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH S MDD without anhedonia MEDRA Medical Dictionary for Regulatory Activities MI Multiple imputation MMRM Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | |
| ICH International Conference on Harmonisation IDMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD Major depressive disorder MDD ANH+ MDD with moderate-to-severe anhedonia MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH S MDD without anhedonia MEDD WOANH S MDD without anhedonia MMRM Mixed model for repeated measures MNAR Missing not at random NSAIDS Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | GI | Gastrointestinal |
| IDMC Independent Data Monitoring Committee IQ Interquartile LS Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD Major depressive disorder MDD ANH+ MDD with moderate-to-severe anhedonia MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MRM Mixed model for repeated measures MNAR Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | HSI | Health status index |
| IQ Interquartile LS Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD Major depressive disorder MDD ANH+ MDD with moderate-to-severe anhedonia MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MCI MED WOANH S MOD without anhedonia MCI MED WOANH S MOD without anhedonia MCI MED WOANH S MOD Without anhedonia MCI MED WOANH S MOD Without anhedonia MCI MED WOANH S MOD Without anhedonia MCI | ICH | International Conference on Harmonisation |
| Least squares MADRS Montgomery-asberg depression rating scale MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD Major depressive disorder MDD ANH+ MDD with moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH S MDD without anhedonia MEDD WOANH S MDD without anhedonia MI Multiple imputation MMRM Mixed model for repeated measures MNAR Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PG-S Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | IDMC | Independent Data Monitoring Committee |
| MADRS Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD Major depressive disorder MDD ANH+ MDD with moderate-to-severe anhedonia MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH S MDD without anhedonia MedDRA Medical Dictionary for Regulatory Activities MI Multiple imputation MMRM Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGG-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | IQ | Interquartile |
| MAR Missing at random MCMC Markov chain monte carlo MCT Meaningful change threshold MDD Major depressive disorder MDD ANH+ MDD with moderate-to-severe anhedonia MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH S MDD without anhedonia MedDRA Medical Dictionary for Regulatory Activities MI Multiple imputation MMRM Mixed model for repeated measures MNAR Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | LS | Least squares |
| MCMC Markov chain monte carlo MCT Meaningful change threshold MDD Major depressive disorder MDD ANH+ MDD with moderate-to-severe anhedonia MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MedDRA Medical Dictionary for Regulatory Activities MI Multiple imputation MMRM Mixed model for repeated measures MNAR Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | MADRS | Montgomery-asberg depression rating scale |
| MCMC Markov chain monte carlo MCT Meaningful change threshold MDD Major depressive disorder MDD ANH+ MDD with moderate-to-severe anhedonia MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MDD WOANH S MDD without anhedonia MEDD WOANH S MDD without anhedonia MEDD WOANH S MDD without anhedonia MEDD WOANH S MOD without anhedonia MEDD | MAR | Missing at random |
| MCT Meaningful change threshold MDD Major depressive disorder MDD ANH+ MDD with moderate-to-severe anhedonia MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH S MDD without anhedonia MedDRA Medical Dictionary for Regulatory Activities MI Multiple imputation MMRM Mixed model for repeated measures MNAR Missing not at random NSAIDS Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | MCMC | |
| MDD Major depressive disorder MDD ANH+ MDD with moderate-to-severe anhedonia MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH S MDD without anhedonia MedDRA Medical Dictionary for Regulatory Activities MI Multiple imputation MMRM Mixed model for repeated measures MNAR Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | |
| MDD ANH+ MDD with moderate-to-severe anhedonia MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH S MDD without anhedonia MedDRA Medical Dictionary for Regulatory Activities MI Multiple imputation MMRM Mixed model for repeated measures MNAR Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | |
| MDD ANH- MDD without moderate-to-severe anhedonia MDD WOANH MS MDD without anhedonia MDD WOANH S MDD without anhedonia MedDRA Medical Dictionary for Regulatory Activities MI Multiple imputation MMRM Mixed model for repeated measures MNAR Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | |
| MDD WOANH MS MDD without anhedonia MedDRA Medical Dictionary for Regulatory Activities MI Multiple imputation MMRM Mixed model for repeated measures MNAR Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | |
| MDD WOANH S MDD without anhedonia MedDRA Medical Dictionary for Regulatory Activities MI Multiple imputation MMRM Mixed model for repeated measures MNAR Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | |
| MedDRA Medical Dictionary for Regulatory Activities MI Multiple imputation MMRM Mixed model for repeated measures MNAR Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | MDD without anhedonia CCI |
| MI Multiple imputation MMRM Mixed model for repeated measures MNAR Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | |
| MMRM Mixed model for repeated measures MNAR Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | |
| MNAR Missing not at random NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | |
| NSAIDs Non-steroidal anti-inflammatory drugs non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | · |
| non-PAP Non primary analysis population PGI-C Physician Global Impression-Change PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | |
| PGI-C Physician Global Impression-Change PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | |
| PGI-S Physician Global Impression-Severity PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | |
| PHQ-9 Patient Health Questionnaire-9 Item PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | |
| PK Pharmacokinetic(s) PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | |
| PWC-20 Physician Withdrawal Checklist 20-items QLDS Quality of life in depression scale | | |
| QLDS Quality of life in depression scale | | V |
| · | | |
| ROW Rest of the world | | |
| | ROW | Rest of the world |

| SAE | Serious adverse event |
|--------|----------------------------------------------|
| SAP | Statistical analysis plan |
| SD | Standard deviation |
| SE | Standard error |
| SHAPS | Snaith-Hamilton Pleasure Scale |
| SMQ | Standardized MedDRA Query |
| SNRI | Selective norepinephrine reuptake inhibitors |
| SSRI | Selective serotonin reuptake inhibitor |
| TE | Treatment emergent |
| WHO-DD | World health organization drug dictionary |

# 6.2. Appendix 2 Changes to Protocol-Planned Analyses

The analysis of exploratory endpoints on the MDD ANH- population (now referred to as non-PAP) stated in the protocol will not be performed as this population contains participants with prominent anhedonia However, these participants will be included in the All MDD population.

## 6.3. Appendix 3 Demographics and Baseline Characteristics

The number of participants in each analysis set will be summarized and listed by intervention group and overall. In addition, the distribution of participants by region, country/territory, and site ID will be presented unless otherwise noted.

Table 7 presents a list of the demographic variables that will be summarized by intervention group and overall for the FAS\_ANH+, MDD\_WOANH\_S, MDD\_WOANH\_MS and safety analysis sets.

**Table 7: Demographic Variables** 

| Continuous Variables | Summary Type |
|---|---|
| Age (years) | Descriptive statistics (N, |
| Weight (kg) | mean, standard deviation |
| Height (cm) | [SD], median and range |
| Body Mass Index (BMI) (kg/m <sup>2</sup> ) | [minimum and maximum]). |
| Categorical Variables | |
| Age group: 18-44, 45-64, 65-74 | |
| Sex (male, female, unknown, undifferentiated) | |
| Race <sup>a</sup> (American Indian or Alaska Native, Asian, Black or African<br>American, Native Hawaiian or other Pacific Islander, White,<br>Multiple, Not Reported) | Frequency distribution with the number and percentage |
| Ethnicity (Hispanic or Latino, not Hispanic or Latino, Not Reported, Unknown) | of participants in each category. |
| Country/territory | |
| Region (South America, North America, Europe, Asia, other) | |
| BMI (underweight <18.5 kg/m², normal 18.5-<25 kg/m², overweight 25-<30 kg/m², obese 30-<40 kg/m², obese >=40 kg/m²) | |
| Employment status (any type of employement, any type of unemployment, other) <sup>b</sup> | |

<sup>&</sup>lt;sup>a</sup> If multiple race categories are indicated, the Race is recorded as 'Multiple'

Table 8 presents a list of the baseline disease characteristics variables that will be summarized by intervention group and overall for the FAS\_ANH+, MDD\_WOANH\_S, MDD\_WOANH\_MS and safety analysis sets.

**Table 8: Psychiatric History at Baseline** 

<sup>&</sup>lt;sup>b</sup> Any type of employment includes: any category containing "Employed", Sheltered Work, Housewife or Dependent Husband, and Student; any type of unemployment includes: any category containing "Unemployed"; Other includes: Retired and No Information Available.

| Continuous Variables | Summary Type |
|---|---|
| Age (years) when diagnosed with MDD | Descriptive statistics |
| Duration (weeks) of current depressive episode | (N, mean, standard |
| Baseline MADRS total score | deviation [SD], |
| Baseline SHAPS total score | median and range |
| Baseline DARS total score | [minimum and |
| Baseline CGI-S score | maximum]). |
| Baseline PGI-S score: anhedonia | |
| Baseline PGI-S score: depression | |
| Baseline PHQ-9 total score | |
| Baseline HDRS-17 total score | |
| Categorical Variables | |
| Number of major depressive episodes (1, 2-5, 6-10, >10) | Frequency |
| Current antidepressant type (SSRI/SNRI) | distribution |
| Number of previous prior antidepressants $(0, 1, 2, 3, >3)$ | with the number and |
| Number of classes of previous ADs received prior to the current AD | percentage of |
| Presence of Medical History (Yes, No) | participants in |
| Baseline CGI-S score (Normal (not at all ill), Borderline mentally ill, Mildly ill, Moderately ill, Markedly ill, Severely ill, Among the most extremely ill patients) | each category. |
| Screening C-SSRS category (no event, suicidal ideation, suicidal behavior) | |
| SCID-CT DSM-5 MDD specifiers for MDD | |
| CCI | |
| Baseline PGI-S score: anhedonia (None, Mild, Moderate, Severe, Very severe) | |
| Baseline PGI-S score: depression (None, Mild, Moderate, Severe, Very severe) | |
| Overall Severity of Anhedonia | |
| Mild | |
| Moderate | |
| Severe | |
| Very severe | |
| Family history of | |
| Alcohol Abuse (Yes, No) | |
| Anxiety Disorder (Yes, No) | |
| Bipolar Disorder (Yes, No) | |
| Depression (Yes, No) | |
| Schizophrenia (Yes, No) | |
| Substance Abuse (Yes, No) | |
| Tabacco usage (Yes, No) | |

<sup>\*</sup> Clinician's assessment of severity of anhedonia is based on clinical evaluation and judgment of impact on the anhedonia domains: interest, motivation, engagement/effort and enjoyment/pleasure.

#### 6.4. Appendix 4 Protocol Deviations

In general, the following list of major protocol deviations may have the potential to impact participants' rights, safety or well-being, or the integrity and/or result of the clinical study. Participants with major protocol deviations will be identified prior to database lock and the participants with major protocol deviations will be summarized by category for FAS\_ANH+ and safety analysis sets.

- Developed withdrawal criteria but not withdrawn
- Entered but did not satisfy criteria
- Received a disallowed concomitant treatment
- Received wrong treatment or incorrect dose
- Other

Number of participants not meeting inclusion criteria, or meeting exclusion criteria will be summarized by study intervention group for the safety analysis set.

If deemed necessary, additional analyses of protocol deviations for assessing and mitigating the impact of COVID-19 on study outcome will be conducted as presented in Appendix 9.

#### 6.5. Appendix 5 Prior and Concomitant Medications

Prior medications and concomitant medications will be coded using the World Health Organization Drug Dictionary (WHO-DD). Prior medications are defined as any therapy used before the day of first dose (partial or complete) of study intervention. Concomitant medications are defined as any therapy used on or after the same day as the first dose of study intervention, including those that started before and continue on after the first dose of study intervention.

Summaries of concomitant medications will be presented by ATC level 2 and level 4 terms and base preferred term for the double-blind and follow-up phases for safety and follow-up analysis sets, respectively. The proportion of participants who receive each concomitant medication will be summarized as well as the proportion of participants who receive at least 1 concomitant medication. In addition, concomitant medications of special interest will be summarized. See Appendix 6 Medications of Special Interest for list of categories of medications of special interest.

Prior antidepressant medications, prior medications other than antidepressants, and prior medications of special interest will be summarized by ATC level 2 and level 4 terms and base preferred term.

# 6.6. Appendix 6 Medications of Special Interest

Categories for medications of special interest are defined as follows:

| Medications of Special Interest Category |
|------------------------------------------------|
| Antidepressants |
| Hypnotic/sedative including z-drugs |
| CCI |
| Non-steroidal anti-inflammatory drugs (NSAIDs) |
| Medications for treatment of CCI |
| Medications for treatment of CCI |

# 6.7. Appendix 7 Conversion of Raw Score to T-Score for PROMIS

| aw Score | Scale Score | SE* |
|----------|-------------|-----|
| 8 | 25.9 | 3.9 |
| 9 | 29.7 | 2.3 |
| 10 | 31.3 | 1.9 |
| 11 | 32.6 | 1.7 |
| 12 | 33.6 | 1.6 |
| 13 | 34.5 | 1.6 |
| 14 | 35.3 | 1.5 |
| 15 | 36.2 | 1.5 |
| 16 | 36.9 | 1.5 |
| 17 | 37.7 | 1.5 |
| 18 | 38.5 | 1.5 |
| 19 | 39.3 | 1.6 |
| 20 | 40.2 | 1.6 |
| 21 | 41.1 | 1.6 |
| 22 | 42.0 | 1.7 |
| 23 | 43.0 | 1.7 |
| 24 | 44.0 | 1.7 |
| 25 | 45.0 | 1.7 |
| 26 | 46.0 | 1.6 |
| 27 | 47.0 | 1.6 |
| 28 | 48.0 | 1.6 |
| 29 | 48.9 | 1.6 |
| 30 | 49.9 | 1.6 |
| 31 | 50.8 | 1.6 |
| 32 | 51.7 | 1.6 |
| 33 | 52.7 | 1.6 |
| 34 | 53.6 | 1.6 |
| 35 | 54.6 | 1.6 |
| 36 | 55.7 | 1.6 |
| 37 | 56.8 | 1.7 |
| 38 | 58.2 | 2.0 |
| 39 | 60.2 | 2.5 |
| 40 | 65.4 | 4.9 |

Adult version

# 6.8. Appendix 8 Criteria for Treatment-emergent Markedly Abnormal Laboratory Values

| Laboratory Parameter | Unit | Low | High |
|---|---|---|---|
| Clinical Chemistry | | | |
| Albumin | g/dL | 2.4 | 6.0 |
| Albumin | g/L | 24 | 60 |
| Alkaline phosphatase | U/L | N/A | 250 |
| Alanine transaminase (SGPT) | U/L | N/A | 200 |
| Aspartate transaminase (SGOT) | U/L | N/A | 250 |
| Bicarbonate | mEq/L | 15.1 | 34.9 |
| Bicarbonate | mmol/L | 15.1 | 34.9 |
| Bilirubin (direct) | mg/dL | N/A | 3.0 |
| Bilirubin (direct) | μmol/L | N/A | 51.3 |
| Bilirubin (total) | mg/dL | N/A | 3.0 |
| Bilirubin (total) | μmol/L | N/A | 51.3 |
| Blood urea nitrogen | mg/dL | N/A | 50 |
| Blood urea nitrogen | mmol/L | N/A | 17.9 |
| Calcium | mg/dL | 6 | 12 |
| Calcium | mmol/L | 1.497 | 2.994 |
| Chloride | mEq/L or mmol/L | 94 | 112 |
| Cholesterol | mg/dL | N/A | 300 |
| Cholesterol | mmol/L | N/A | 7.758 |
| Creatine kinase | U/L | N/A | 990 |
| Creatinine | mg/dL | N/A | 3 |
| Creatinine | μmol/L | N/A | 265.2 |
| Gamma glutamyl transferase | U/L | N/A | 300 |
| Glucose Plasma | mg/Dl | 40 | 300 |
| Glucose Plasma | mmol/L | 2.204 | 16.653 |
| Hemoglobin A1c | Fraction of 1 | 0.04 | 0.08 |
| High-density lipoprotein cholesterol (HDL) | mg/dL | 35 | N/A |
| High-density lipoprotein cholesterol (HDL) | mmol/L | 0.905 | N/A |
| Low-density lipoprotein cholesterol (LDL) | mg/dL | 89 | 160 |
| Low-density lipoprotein cholesterol (LDL) | mmol/L | 2.3015 | 4.1376 |
| Phosphate | mg/dL | 2.2 | 8.1 |
| Phosphate | mmol/L | 0.71038 | 2.61549 |
| Potassium | mmol/L | 3.0 | 5.8 |
| Sodium | mEq/L | 125 | 155 |
| Sodium | mmol/L | 125 | 155 |
| Total protein | g/L | 50 | N/A |
| Triglycerides | mg/dL | N/A | 500 |
| Triglycerides | mmol/L | N/A | 5.645 |
| Uric acid | mg/dL | 1.5 | 10 |
| Uric acid | μmol/L | 89.22 | 594.8 |
| Hematology | | | |
| Hematocrit - female | % | 0.28 | 0.50 |

CONFIDENTIAL – FOIA Exemptions Apply in U.S. Status: Approved, Date: 03 October 2024

| - male | % | 0.24 | 0.55 |
|---|---|---|---|
| Hemoglobin | g/dL | 8 | 19 |
| Hemoglobin | g/L | 80 | 190 |
| Neutrophils | % | 30 | 90 |
| Monocytes | % | N/A | 20 |
| Eosinophils | % | N/A | 10 |
| Basophils | % | N/A | 6 |
| Lymphocytes | % | 10 | 60 |
| Reticulocytes | % | 0.5 | 1.5 |
| Platelet count | 10 <sup>9</sup> /L; giga/L | 100 | 600 |
| Red blood cell (RBC) count - female | 10 <sup>12</sup> /L; tera/L | 3.0 | 5.5 |
| - male | 10 <sup>12</sup> /L; tera/L | 3.0 | 6.4 |
| White blood cell (WBC) count | 10 <sup>9</sup> /L; giga/L | 2.5 | 15.0 |
| Urinalysis | | | |
| Urine pH | | N/A | 6.5 |
| Urine specific gravity | | < 1.001 | > 1.035 |

Note: Values should be flagged as markedly abnormally low if the value is less than the value indicated in the "Low" column. Likewise, values should be flagged as markedly abnormally high if the value is greater than the value indicated in the "High" column.

Note: The same limits apply to both males and females unless gender is indicated.

N/A = Not applicable

## 6.9. Appendix 9 Analyses for Assessing and Mitigating the Impact of COVID-19 on Study Outcome

The following measures will be taken to handle the impact of COVID-19 on study outcome:

- 1. Listing and summary of treatment discontinuation and study discontinuation including reasons due to COVID-19 will be presented.
- 2. Protocol deviation related to COVID-19 including missing visits and remote visits due to COVID will be summarized; corresponding listing will be provided.
- 3. Additional analyses to assess the potential impact of COVID-19 in the primary and key secondary endpoints.
  - a. Mean summaries over time by types of collection (remote, home, site, etc).
  - b. Sensitivity analyses will be provided by including types of collection in the primary models for MADRS and DARS.
- 4. Sensitivity analysis for the primary Estimand ROW: Additional tipping point analysis will be performed for the primary Estimand ROW where the delta adjustments will be applied to missing data under hypothetical strategy including those caused by discontinuation reasons due to COVID- 19; delta adjustments will not be applied to data due to discontinuation reasons not related to study intervention including Lost to Follow-Up, Withdrawal by Subject or Other.

Note: The above measures will be taken in instances where a large number of COVID infections are reported. A few isolated cases of COVID-19 infection reported by the participants will not warrant the above analyses.

## 6.10. Appendix 10 Delta Adjustment Multiple Imputation

1. If the data has non-monotone missing data, then impute any intermediate missing data with Markov Chain Monte Carlo method.

```
/*visits v1-v3 are corresponding to Day 15, 29 and 43 for MADRS, trt=2 is for control group*/
  proc mi data=MADRS data nimpute=500 seed=1234 out=MADRS mcmc noprint;
    var treatment baselinecountry/territory v1-v3;
    mcmc chain=single nbiter=200 niter=100 impute=monotone;
  proc sort; by imputation;
  run;
 2. Delta adjustment
 %macro procmib deltamar(indata=,deltac=,deltad=);
    data indata mi;
      set MADRS mcmc:
      v1 mi=v1;v2 mi=v2;v3 mi=v3;
/*Perform MI with monotone regression method*/
/*As multiple datasets have been already created with MCMC, use only nimpute=1*/
/*If original dataset has monotone missing data, use nimpute>1 such as 500*/
    proc mi data=indata mi out=reg nimpute=1 seed=123 noprint;
     by imputation;
      var trt base v1 mi v2 mi v3 mi;
      class trt;
      monotone regression;
    run;
   data regd;
     set reg;
      if trt=1 then do;
        if v1=. then v1 mi=v1 mi-&deltac;
        if v2=. then v2 mi=v2 mi-&deltac;
        if v3=. then v3 mi=v3 mi-&deltac;
      end;
      if trt=2 then do:
       if v1=. then v1 mi=v1 mi+&deltad;
       if v2=. then v2 mi=v2 mi+&deltad;
       if v3=. then v3 mi=v3 mi+&deltad;
      end;
   run;
  data regsd;
      c1 mi=v1 mi-base;c2 mi=v2 mi-base;c3 mi=v3 mi-base;
```

CONFIDENTIAL - FOIA Exemptions Apply in U.S.

proc sort data; by imputation;

```
run;
 %mend;
 %procmib deltamar(indata=MADRS mcmc,deltac=0,deltad=1);
 3. Analyze fully imputed datasets with MMRM
   data MADRS reg subset;
     set regsd;
     keep imputation ID Country trt base c1 mi c2 mi c3 mi;
   proc sort data=MADRS reg subset;
        by ID Country trt base imputation;
    run;
   proc transpose data=MADRS reg subset
                  out=MADRS mi vertical name=visit prefix=change;
         by ID Country trt base imputation;
   run;
   data MADRS mi vertical;
     set MADRS mi vertical;
       rename change1=change;
       if visit="c1 mi" then visitn=1;
       if visit="c2 mi" then visitn=2;
       if visit="c3 mi" then visitn=3;
   proc sort; by imputation ID visitn;
   run;
   proc mixed data=MADRS mi vertical;
           by imputation;
           class trt Country visitn id;
           model change = base trt Country visitn trt*visitn /ddfm=kr;
           repeated visitn / sub = id type = un;
           lsmeans trt*visitn/ diff=control('2' '3');
           ods output lsmeans=lsm mib diffs=diff mib;
    run;
 4. Pool the results with Rubin's rules
   proc mianalyze parms=diffmi;
       class trt visitn;
       model effects treatment; /* check to see what MMRM outputs to determine which
variables to include */
       ods output parameterestimates=diffmian;
```

Status: Approved, Date: 03 October 2024

run;

## 6.11. Appendix 11 AE Suggested to Abuse Potential (PTs)

Potential abuse-related AEs are defined as below:

- SMQ "Drug Abuse, Dependence and Withdrawal"
- SMQ "Psychosis and Psychotic Disorders"
- MedDRA preferred terms (PTs):

Aggression; Confusional state; Decreased activity; Dependence; Disorientation; Dissociation; Dissociative disorder; Dizziness; Drug abuse; Drug abuser; Drug dependence; Drug detoxification; Drug diversion; Drug rehabilitation; Drug tolerance; Drug tolerance increased; Drug use disorder; Drug withdrawal convulsions; Drug withdrawal headache; Drug withdrawal syndrome; Euphoric mood; Feeling abnormal; Feeling drunk; Feeling of relaxation; Hallucination; Hallucination, auditory; Hallucination, gustatory; Hallucination, olfactory; Hallucination, synaesthetic; Hallucination, tactile; Hallucination, visual; Hallucinations, mixed; Inappropriate affect; Mental impairment; Product tampering; Psychomotor hyperactivity; Psychotic disorder; Rebound effect; Somatic hallucination; Somnolence; Substance abuser; Substance dependence; Substance use; Substance use disorder; Substance-induced mood disorder; Substance-induced psychotic disorder; Thinking abnormal; Withdrawal arrhythmia; Withdrawal syndrome

• Standardized MedDRA Query (SMQ) and Custom MedDRA Query (CMQ) analyses:

Dopamine dysregulation syndrome; Drug abuse; Drug abuser; Drug dependence; Drug dependence, antepartum; Drug dependence, postpartum; Drug use disorder; Drug use disorder, antepartum; Drug use disorder, postpartum; Intentional overdose; Intentional product misuse; Maternal use of illicit drugs; Neonatal complications of substance abuse; Substance abuse; Substance abuser; Substance dependence; Substance use disorder; Accidental overdose; Dependence; Disturbance in social behaviour; Drug detoxification; Drug diversion; Drug level above therapeutic; Drug level increased; Drug screen; Drug screen positive; Drug tolerance; Drug tolerance decreased; Drug tolerance increased; Intentional product use issue; Medication overuse headache; Narcotic bowel syndrome; Needle track marks; Overdose; Prescription drug used without a prescription; Prescription form tampering; Reversal of opiate activity; Substance use; Substance-induced mood disorder; Substanceinduced psychotic disorder; Toxicity to various agents; Drug withdrawal convulsions; Drug withdrawal headache; Drug withdrawal maintenance therapy; Drug withdrawal syndrome; Drug withdrawal syndrome neonatal; Drug rehabilitation; Rebound effect; Steroid withdrawal syndrome; Withdrawal arrhythmia; Withdrawal catatonia; Withdrawal syndrome; Behavioural addiction; Intentional device use issue; Anti-androgen withdrawal syndrome; Intentional device misuse; Product administered at inappropriate site; Alcohol use disorder; Performance enhancing product use; Intentional misuse of drug delivery system; Cholinergic rebound syndrome; Steroid dependence; Cannabinoid hyperemesis syndrome; Delusion of parasitosis; Behavioral addiction

Note: Some of the PTs listed above are included in the *Drug Abuse*, *Dependence and Withdrawal*, and *Psychosis and Psychotic Disorders* SMQs

# 6.12. Appendix 12 Spaghetti Plot of MADRS Change Over Time (Study 67953964MDD2001)

Change in MADRS Total Score by Reason for Discontinuation from the Study (MDD2001)



CONFIDENTIAL - FOIA Exemptions Apply in U.S.

# 6.13. Appendix 13 Quality Tolerance Limits (QTLs)

Quality Tolerance Limit (QTL) parameters and thresholds are defined and will be monitored in in this study. QTL parameters will be summarized. More details are described in the Integrated Analytic Risk-Based Monitoring (iARBM) Plan.

# 6.14. Appendix 14 Scoring of QLDS items





#### 7. REFERENCES

- 1. EuroQol Group. About EQ-5D. http://www.euroqol.org/about-eq-5d.html (Accessed 18 Jun 2014).
- 2. EuroQol Group. EQ-5D-5L User Guide: basic information on how to use the EQ-5D-5L instrument. Version 2.0; Oct 2013.
  - http://www.euroqol.org/fileadmin/user\_upload/Documenten/PDF/Folders\_Flyers/UserGuide\_EQ-5D-5L v2.0 October 2013.pdf (Accessed 6 Aug 2014).
- 3. Feng X, Eleanor P etc. A Time Trade-off-derived Value Set of the EQ-5D-5L for Canada. Med Care, 2016 Jan;54(1):98-105
- 4. Franken IH, Rassin E, Muris P. The assessment of anhedonia in clinical and non-clinical populations: further validation of the Snaith-Hamilton Pleasure Scale (SHAPS). J Affect Disord. 2007;99(1-3):83-89.
- 5. Guy W. CGI: Clinical Global Impressions. In: ECDEU Assessment Manual for Psychopharmacology. Rockville, MD: US Department of Health and Human Services; printed 1976 (reprinted 1991):217-222.
- 6. Health Measures (2016). PROMIS Short Form v2.0 Ability to Participate in Social Roles and Activities 8a. Dated 23 June 2016.
- 7. Hunt SM (1992), McKenna SP. The QLDS: as scale for the measurement of quality of life in depression. Health Policy. 1992;22(3):307-319.
- 8. Hunt SM. A new measure of quality of life in depression: testing the reliability and construct validity of the QLDS. Health Policy. 1992;22(3):321-330.
- 9. Imai K, Keele L, Tingley D (2010). A general approach to causal mediation analysis. Psychological Methods, Vol. 15, No. 4, pp. 309–334.
- 10. Imai K, Keele L, Yamamoto T. Identification, Inference, and Sensitivity Analysis for Causal Mediation Effects. Statistical Science, 2010; 25(1), 51–71.
- 11. Investigator's Brochure: JNJ-67953964 (aticaprant), edition 6. Janssen Research & Development (20 Jan 2022)McKenna SP (1992),
- 12. Khin NA. Update on FDA exploratory analyses of aggregated efficacy data from antidepressant trials. Presented at NCDEU Regulatory Plenary. New FDA & EMA initiatives in Alzheimer's disease, depression and schizophrenia. May 30, 2013
- 13. McGahuey CA, Gelenberg AJ, Laukes CA, et al. The Arizona Sexual Experience Scale (ASEX): reliability and validity. J Sex Marital Ther. 2000;26(1):25-40.

- 14. McKenna SP (1992), Hunt SM. A new measure of quality of life in depression: testing the reliability and construct validity of the OLDS. Health Policy. 1992;22(3):321-330.
- 15. Nakonezny PA, Carmody TJ, Morris DW, Kurian BT, Trivedi MH. Psychometric evaluation of the Snaith– Hamilton Pleasure Scale (SHAPS) in adult outpatients with major depressive disorder. Int Clin Psychopharmacol 2010;25(6):328-333.
- 16. Posner K, Oquendo MA, Gould M, Stanley B, Davies M. Columbia Classification Algorithm of Suicide Assessment (C-CASA): classification of suicidal events in the FDA's pediatric suicidal risk analysis of antidepressants. Am J Psychiatry. 2007;164:1035-1043.
- 17. PROMIS Ability to Participate in Social Roles and Activities Scoring Manual: https://www.assessmentcenter.net/ac scoringservice
- 18. Rubin, D. (1987), Multiple Imputation for Nonresponse in Surveys, Wiley, New York, XXIX+258 pp.
- 19. Rizvi SJ, Quilty LC, Sproule BA, Cyriac A, Michael Bagby R, Kennedy SH. Development and validation of the Dimensional Anhedonia Rating Scale (DARS) in a community sample and individuals with major depression. Psychiatry Res. 2015;229(1-2):109-119.
- 20. Snaith RP, Hamilton M, Morley S, Humayan A, Hargreaves D, Trigwell P. A scale for the assessment of hedonic tone the Snaith-Hamilton Pleasure Scale. Br J Psychiatry. 1995;167(1):99-103.
- Siddiqui, Ohidul, HM James Hung, and Robert O'Neill. "MMRM vs. LOCF: a comprehensive comparison based on simulation study and 25 NDA datasets." Journal of biopharmaceutical statistics 19.2 (2009): 227-246.
- 22. Spitzer RL (1999), Kroenke K, Williams JB. Validation and utility of a self-report version of PRIME-MD: the PHQ primary care study. JAMA. 1999;282:1737-1744.
- 23. Spitzer RL (2006), Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006;166(10):1092-1097.
- 24. Tingley, D., Yamamoto, T., Hirose, K., Keele, L., & Imai, K. Mediation: R Package for Causal Mediation Analysis. Journal of Statistical Software, 2014; 59(5), 1–38. https://doi.org/10.18637/jss.v059.i05
- 25. Tuynman-Qua H (1997), de Jonghe F, McKenna SP. Quality of life in depression scale (QLDS). Development, reliability, validity, responsiveness and application. Eur Psychiatry. 1997;12(4):199-202.
- 26. Yang P (2013). Recent advances in design and methodology in psychiatric clinical trials. Presented at: Joint Statistical Meetings, Montréal, QC Canada, August 3-8, 2013
- 27. VanderWeele TJ. Explanation in Causal Inference: Methods for Mediation and Interaction. New York, NY: Oxford University Press. 2015.